CLINICAL TRIAL: NCT03632720
Title: Immunogenicity and Safety Study of an Investigational Quadrivalent Meningococcal Conjugate Vaccine in Infants and Toddlers When Administered Using a 1+1 Schedule in a National Immunization Schedule Having a Meningococcal Group B Vaccine as Standard of Care
Brief Title: Immunogenicity and Safety of a Quadrivalent Meningococcal Conjugate Vaccine in Infants and Toddlers When Administered Concomitantly With Routine Pediatric Vaccines in the United Kingdom
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MET52; 2017-004520-30 (EudraCT Number); U1111-1183-6530 (Registry Identifier: ICTRP)
Record Dates: First submitted 2018-08-03; First posted 2018-08-15 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers (Meningococcal Infection)
MeSH Terms: conditions — Meningococcal Infections | interventions — 4CMenB vaccine; Tetanus Toxoid; Hepatitis B Vaccines; Vaccines; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; RIX4414 vaccine; 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) (Experimental): Participants aged 2 months (at the time of enrollment) received MenACYW Conjugate vaccine at 3 months and at 12 to 13 months of age, Bexsero® at 2, 4, and 12 to 13 months of age along with Infanrix hexa® vaccine at 2, 3, and 4 months of age; Rotarix® vaccine at 2 and 3 months of age; and Prevenar 13® vaccine at 2 and 4 months of age.
  Interventions: Biological: Meningococcal polysaccharide (serogroups A,C,Y and W) tetanus toxoid Conjugate vaccine; Biological: Meningococcal group B vaccine; Biological: Diphtheria, tetanus, pertussis (acellular component), hepatitis B, poliomyelitis (inactivated) vaccine; Biological: Human rotavirus RIX4414 strain vaccine; Biological: Pneumococcal 13-valent polysaccharide conjugate vaccine
- Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months) (Experimental): Participants aged 2 months (at the time of enrollment) received MenACYW Conjugate vaccine at 3 months and at 12 to 13 months of age, Bexsero® at 2 and 4 months of age along with Infanrix hexa® vaccine at 2, 3, and 4 months of age; Rotarix® vaccine at 2 and 3 months of age; and Prevenar 13® vaccine at 2 and 4 months of age.
  Interventions: Biological: Meningococcal polysaccharide (serogroups A,C,Y and W) tetanus toxoid Conjugate vaccine; Biological: Meningococcal group B vaccine; Biological: Diphtheria, tetanus, pertussis (acellular component), hepatitis B, poliomyelitis (inactivated) vaccine; Biological: Human rotavirus RIX4414 strain vaccine; Biological: Pneumococcal 13-valent polysaccharide conjugate vaccine
- Group 3: Bexsero® (2, 4, and 12 to 13 Months) (Active Comparator): Participants aged 2 months (at the time of enrollment) received Bexsero® at 2, 4, and 12 to 13 months of age along with Infanrix hexa® vaccine at 2, 3, and 4 months of age; Rotarix® vaccine at 2 and 3 months of age; and Prevenar 13® vaccine at 2 and 4 months of age.
  Interventions: Biological: Meningococcal group B vaccine; Biological: Diphtheria, tetanus, pertussis (acellular component), hepatitis B, poliomyelitis (inactivated) vaccine; Biological: Human rotavirus RIX4414 strain vaccine; Biological: Pneumococcal 13-valent polysaccharide conjugate vaccine

INTERVENTIONS:
Biological: Meningococcal polysaccharide (serogroups A,C,Y and W) tetanus toxoid Conjugate vaccine — Pharmaceutical form: solution for injection; route of administration: intramuscular, 0.5 mL
  Other Names: MenACYW Conjugate vaccine
  Arms: Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months); Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Biological: Meningococcal group B vaccine — Pharmaceutical form: suspension for injection; route of administration: deep intramuscular, 0.5 mL
  Other Names: Bexsero®
Biological: Diphtheria, tetanus, pertussis (acellular component), hepatitis B, poliomyelitis (inactivated) vaccine — Pharmaceutical form: powder and suspension for suspension injection; route of administration: deep intramuscular, 0.5 mL
  Other Names: Infanrix hexa®
Biological: Human rotavirus RIX4414 strain vaccine — Pharmaceutical form: oral suspension; route of administration: oral, 1.5 mL
  Other Names: Rotarix®
Biological: Pneumococcal 13-valent polysaccharide conjugate vaccine — Pharmaceutical form: suspension for injection; route of administration: intramuscular, 0.5 mL
  Other Names: Prevenar 13®

SUMMARY:
The primary objective of the study was to demonstrate the non-inferiority of the antibody responses to meningococcal serogroups A, C, W, and Y (MenACYW) in terms of serum bactericidal assay using human complement (hSBA) vaccine seroprotection (antibody titer greater than or equal to [>=] 1:8) when MenACYW Conjugate vaccine was administered concomitantly with Bexsero® in the second year of life compared to when MenACYW Conjugate vaccine was given alone.

The secondary objectives were to compare the hSBA antibody response in terms of geometric mean titers (GMTs) against meningococcal serogroups A, C, W, and Y when MenACYW Conjugate vaccine was administered concomitantly with Bexsero® or when MenACYW Conjugate vaccine was given alone in the second year of life; to describe the hSBA and serum bactericidal assay using baby rabbit complement (rSBA) antibody responses against meningococcal serogroups A, C, W, and Y before and after the 1st dose of MenACYW Conjugate vaccine administered at 3 months of age, before and after the 2nd dose of MenACYW Conjugate vaccine administered at 12 to 13 months of age for Group 1 and Group 2; to describe the hSBA and rSBA antibody persistence against meningococcal serogroups A, C, W, and Y after the 1st dose of MenACYW Conjugate vaccine administered at 3 months of age for Group 1 and Group 2.

DETAILED DESCRIPTION:
Study duration per participant was approximately 11 to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged >= 56 to less than or equal to (<=) 89 days on the day of the first study visit.
* Born at full term of pregnancy (>= 37 weeks) and with a birth weight >= 2.5 kilogram (kg) (or 5 lb and 8 oz).
* Informed consent form had been signed and dated by the parent(s) or other legally acceptable representative (and by an independent witness if required by local regulations).
* Participant and parent/legally acceptable representative were able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

-- Participation at the time of study enrollment (or in the 4 weeks preceding the first trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.

* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination (at Visit 1) or planned receipt of any vaccine in the 4 weeks before and/or following any trial vaccination except for influenza vaccination, which may be received at a gap of at least 2 weeks before or 2 weeks after any study vaccines. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines.
* Previous vaccination against meningococcal disease with either the trial vaccine or another vaccine (i.e., mono- or polyvalent, polysaccharide, or conjugate meningococcal vaccine containing serogroups A, C, W, or Y; or meningococcal B serogroup-containing vaccine).
* Previous vaccination (before Visit 1) with any pneumococcal, diphtheria, tetanus, pertussis, hepatitis B, Haemophilus influenzae type b (Hib), poliovirus, and/or rotavirus vaccines. Receipt of BCG vaccine at birth was acceptable.
* Receipt of immune globulins, blood or blood-derived since birth.
* Known or suspected congenital or acquired immunodeficiency, including Severe Combined Immunodeficiency disorder (SCID); or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks) since birth.
* History of any neurologic disorders, including any seizures and progressive neurologic disorders or encephalopathy.
* History of Neisseria meningitidis infection, confirmed either clinically, serologically, or microbiologically.
* History of diphtheria, tetanus, pertussis, poliomyelitis, Hib, hepatitis B, Streptococcus pneumoniae, and/or rotavirus infection or disease.
* At high risk for meningococcal infection during the trial (specifically, but not limited to, participants with persistent complement deficiency, with anatomic or functional asplenia, or participants travelling to countries with high endemic or epidemic disease).
* History of Guillain-Barré syndrome.
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances including neomycin, kanamycin, polymyxin, formaldehyde, and latex.
* Hereditary problems of fructose intolerance, glucose-galactose malabsorption or sucrase-isomaltase insufficiency.
* History of intussusception or uncorrected congenital malformation of the gastrointestinal tract that would predispose to intussusception.
* Verbal report of thrombocytopenia, contraindicating intramuscular vaccination in the investigator's opinion.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination.
* Chronic illness that, in the opinion of the investigator, was at a stage where it might interfere with trial conduct or completion.
* Any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives, including planning to leave the area of the study site before the end of the study.
* Moderate or severe acute illness/infection (according to investigator judgment), or febrile illness (temperature >= 38.0°C), or diarrhea or vomiting on the day of vaccination. A prospective participant should not be included in the study until the condition had resolved or the febrile event has subsided.
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study.

Ages: 56 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 788 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (13):
- United Kingdom (13):
  - Investigational Site Number :8260024, Newquay, Cornwall
  - Investigational Site Number :8260009, Penzance, Cornwall
  - Investigational Site Number :8260013, Torpoint, Cornwall
  - Investigational Site Number :8260010, Exeter, Devon
  - Investigational Site Number :8260017, Poole, Dorset
  - Investigational Site Number :8260018, Gloucester, Gloucestershire
  - Investigational Site Number :8260001, Bristol
  - Investigational Site Number :8260011, Ivybridge
  - Investigational Site Number :8260002, London
  - Investigational Site Number :8260004, Manchester
  - Investigational Site Number :8260003, Southampton
  - Investigational Site Number :8260006, Taunton
  - Investigational Site Number :8260021, Waterlooville

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 16 sites in United Kingdom from 10 October 2018 to 05 December 2022.
Pre-assignment Details: A total of 788 participants were enrolled and randomized in the study.
Groups:
- Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months): Participants aged 2 months (at the time of enrollment) received Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus toxoid (MenACYW) Conjugate vaccine at 3 months and at 12 to 13 months of age, Bexsero® at 2, 4, and 12 to 13 months of age along with Infanrix hexa® vaccine at 2, 3, and 4 months of age; Rotarix® vaccine at 2 and 3 months of age; and Prevenar 13® vaccine at 2 and 4 months of age.
Period: Overall Study
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months) | Group 3: Bexsero® (2, 4, and 12 to 13 Months)
Started | 314 | 316 | 158
Safety Analysis Set (Safety analysis set included all participants who had received at least 1 dose of study vaccines and had any safety data available. All participants had their safety analyzed after each dose according to the vaccine they actually received at each visit, and after any dose according to the vaccine received.) | 314 | 314 | 157
Completed | 301 | 305 | 150
Not Completed | 13 | 11 | 8
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by parent/legally acceptable representative | 11 | 9 | 8
Not completed — Screen failure | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months) | Group 3: Bexsero® (2, 4, and 12 to 13 Months) | Total
Number analyzed (Participants) | 314 | 316 | 158 | 788
Age, Continuous [Mean (Standard Deviation); unit: days] | 64.7 (6.88) | 63.9 (6.73) | 64.8 (7.03) | 64.4 (6.85)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 166 | 161 | 77 | 404
  Female | 148 | 154 | 81 | 383
  Missing | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 4 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 300 | 296 | 148 | 744
  More than one race | 4 | 10 | 4 | 18
  Unknown or Not Reported | 9 | 4 | 2 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Antibody Titers Greater Than or Equal to (>=) 1:8 Against Meningococcal Serogroups A, C, Y, and W Measured by hSBA After Vaccination: Groups 1 and 2 - PPAS3
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by serum bactericidal assay using human complement (hSBA) assay. Percentage of participants with antibody titers >=1:8 for meningococcal serogroups A, C, Y, and W were reported in this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for Group 3.
Time Frame: 30 days post-vaccination at the age of 12 to 13 months (i.e., at the age of 13 to 14 months)
Population: Analysis was performed on Per-Protocol Analysis Set 3 (PPAS3) defined for accessing ACYW immune response data for participants who received at least 1 dose of study vaccine and had valid post-vaccination serology results of 2nd year of life, with no relevant protocol deviation. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 178 | 169
percentage of participants
  Serogroup A: number analyzed (Participants) | 159 | 156
  Serogroup A | 100 [97.7 to 100] | 99.4 [96.5 to 100]
  Serogroup C: number analyzed (Participants) | 168 | 165
  Serogroup C | 100 [97.8 to 100] | 100 [97.8 to 100]
  Serogroup Y: number analyzed (Participants) | 161 | 159
  Serogroup Y | 100 [97.7 to 100] | 100 [97.7 to 100]
  Serogroup W: number analyzed (Participants) | 172 | 160
  Serogroup W | 99.4 [96.8 to 100] | 100 [97.7 to 100]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) vs Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months); Serogroup A; Test type: Non-Inferiority — The overall non-inferiority was demonstrated if the lower limit of the 2-sided 95 percent (%) confidence interval (CI) was greater (>) -10% for all four serogroups; Difference in Percentage = 0.64, 95% CI 2-sided [-1.78 to 3.54]
Statistical Analysis 2: Comparison: Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) vs Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months); Serogroup C; Test type: Non-Inferiority — The overall non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI was > -10% for all four serogroups; Difference in Percentage = 0.00, 95% CI 2-sided [-2.24 to 2.28]
Statistical Analysis 3: Comparison: Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) vs Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months); Serogroup Y; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in Percentage = 0.00, 95% CI 2-sided [-2.33 to 2.36]
Statistical Analysis 4: Comparison: Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) vs Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months); Serogroup W; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in Percentage = -0.58, 95% CI 2-sided [-3.22 to 1.81]

2. Secondary Outcome: Geometric Mean Titers (GMTs) of Antibodies Measured by hSBA Against Meningococcal Serogroups A, C, Y, and W After Vaccination: Group 1 and 2 - PPAS3
Description: GMTs of antibody against meningococcal serogroups A, C, Y, and W were measured by hSBA. Titers were expressed in terms of 1/dilution.
Time Frame: 30 days post-vaccination at the age of 12 to 13 months (i.e., at the age of 13 to 14 months)
Population: Analysis was performed on PPAS3. Here, 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for Group 3.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 178 | 169
titers
  Serogroup A: number analyzed (Participants) | 159 | 156
  Serogroup A | 1214 [993 to 1484] | 205 [168 to 250]
  Serogroup C: number analyzed (Participants) | 168 | 165
  Serogroup C | 963 [784 to 1182] | 744 [608 to 911]
  Serogroup Y: number analyzed (Participants) | 161 | 159
  Serogroup Y | 454 [374 to 551] | 434 [359 to 525]
  Serogroup W: number analyzed (Participants) | 172 | 160
  Serogroup W | 578 [478 to 698] | 528 [439 to 635]

3. Secondary Outcome: Geometric Mean Titers of Antibodies Measured by hSBA Against Meningococcal Serogroups A, C, Y, and W Before Vaccination: Group 1 and 2 - PPAS1
Description: GMTs of antibody against meningococcal serogroups A, C, Y, and W were measured by hSBA. Infancy was defined as up to 4 months of age. Titers were expressed in terms of 1/dilution. Data for this outcome measure was not planned to be collected and analyzed for Group 3.
Time Frame: Before vaccination at the age of 3 months
Population: Analysis was performed on per-protocol analysis set 1 (PPAS1) defined for accessing ACYW immune response data for participants who received at least 1 dose of study vaccine and had valid post-vaccination serology result of infancy (up to 4 months age) vaccination stage, with no relevant protocol deviations. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 78 | 77
titers
  Serogroup A: number analyzed (Participants) | 22 | 27
  Serogroup A | 8.52 [5.16 to 14.1] | 7.22 [4.39 to 11.9]
  Serogroup C: number analyzed (Participants) | 27 | 34
  Serogroup C | 3.70 [2.84 to 4.84] | 3.84 [2.49 to 5.92]
  Serogroup Y: number analyzed (Participants) | 27 | 30
  Serogroup Y | 3.26 [2.23 to 4.76] | 2.58 [2.17 to 3.07]
  Serogroup W: number analyzed (Participants) | 24 | 29
  Serogroup W | 2.52 [1.93 to 3.30] | 2.15 [1.98 to 2.33]

4. Secondary Outcome: Geometric Mean Titers of Antibodies Measured by hSBA Against Meningococcal Serogroups A, C, Y, and W After Vaccination: Group 1 and 2 - PPAS1
Description: as for outcome 3
Time Frame: 30 days post-vaccination at the age of 3 months (i.e., at the age of 4 months)
Population: Analysis was performed PPAS1. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 78 | 77
titers
  Serogroup A: number analyzed (Participants) | 64 | 71
  Serogroup A | 10.8 [8.40 to 14.0] | 9.63 [7.46 to 12.4]
  Serogroup C: number analyzed (Participants) | 77 | 77
  Serogroup C | 78.0 [52.9 to 115] | 61.2 [41.3 to 90.7]
  Serogroup Y: number analyzed (Participants) | 71 | 68
  Serogroup Y | 9.44 [7.16 to 12.5] | 6.33 [4.93 to 8.13]
  Serogroup W: number analyzed (Participants) | 76 | 73
  Serogroup W | 4.67 [3.74 to 5.83] | 3.81 [3.12 to 4.66]

5. Secondary Outcome: Geometric Mean Titers of Antibodies Measured by hSBA Against Meningococcal Serogroups A, C, Y, and W Before Vaccination: Group 1 and 2 - PPAS3
Description: GMTs of antibodies against meningococcal serogroups A, C, Y, and W were measured by hSBA. Infancy was defined as up to 4 months of age. Titers were expressed in terms of 1/dilution.
Time Frame: Before vaccination at the age of 12 to 13 months
Population: Analysis was performed on PPAS3. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for Group 3.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 35 | 26
titers
  Serogroup A: number analyzed (Participants) | 31 | 26
  Serogroup A | 45.8 [28.4 to 73.8] | 22.6 [13.5 to 37.9]
  Serogroup C | 30.2 [19.0 to 47.9] | 8.44 [5.18 to 13.7]
  Serogroup Y: number analyzed (Participants) | 32 | 26
  Serogroup Y | 25.2 [16.8 to 37.8] | 9.90 [6.43 to 15.3]
  Serogroup W | 34.6 [21.4 to 56.1] | 10.4 [6.58 to 16.6]

6. Secondary Outcome: Geometric Mean Titers of Antibodies Measured by hSBA Against Meningococcal Serogroups A, C, Y, and W After Vaccination: Group 1 and 2 - PPAS3
Description: GMTs of antibodies against meningococcal serogroups A, C, Y, and W were measured by hSBA. Titers were expressed in terms of 1/dilution.
Time Frame: 30 days post-vaccination at the age of 12 to 13 months (i.e., at the age of 13 to 14 months)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 178 | 169
titers
  Serogroup A: number analyzed (Participants) | 159 | 156
  Serogroup A | 1214 [993 to 1484] | 205 [168 to 250]
  Serogroup C: number analyzed (Participants) | 168 | 165
  Serogroup C | 963 [784 to 1182] | 744 [608 to 911]
  Serogroup Y: number analyzed (Participants) | 161 | 159
  Serogroup Y | 454 [374 to 551] | 434 [359 to 525]
  Serogroup W: number analyzed (Participants) | 172 | 160
  Serogroup W | 578 [478 to 698] | 528 [439 to 635]

7. Secondary Outcome: Geometric Mean Titers of Antibodies Measured by rSBA Against Meningococcal Serogroups A, C, Y, and W Before Vaccination: Group 1 and 2 - PPAS1
Description: GMTs of antibodies against meningococcal serogroups A, C, Y, and W were measured by serum bactericidal assay using baby rabbit complement (rSBA). Infancy was defined as up to 4 months of age. Titers were expressed in terms of 1/dilution.
Time Frame: Before vaccination at the age of 3 months
Population: Analysis was performed on PPAS1. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for Group 3.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 47 | 51
titers
  Serogroup A: number analyzed (Participants) | 16 | 22
  Serogroup A | 2.00 [NA to NA] — 95% confidence interval (CI) was not computable as the standard deviation (SD) of the sample was 0, since all participants had the same value. | 2.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value.
  Serogroup C: number analyzed (Participants) | 19 | 23
  Serogroup C | 2.88 [1.84 to 4.52] | 3.77 [2.01 to 7.04]
  Serogroup Y: number analyzed (Participants) | 19 | 23
  Serogroup Y | 2.68 [1.76 to 4.08] | 2.70 [1.87 to 3.92]
  Serogroup W: number analyzed (Participants) | 17 | 23
  Serogroup W | 2.89 [1.69 to 4.94] | 2.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value.

8. Secondary Outcome: Geometric Mean Titers of Antibodies Measured by rSBA Against Meningococcal Serogroups A, C, Y, and W After Vaccination: Group 1 and 2 - PPAS1
Description: GMTs of antibodies against meningococcal serogroups A, C, Y, and W were measured by rSBA. Infancy was defined as up to 4 months of age. Titers were expressed in terms of 1/dilution.
Time Frame: 30 days post-vaccination at the age of 3 months (i.e., at the age of 4 months)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 47 | 51
titers
  Serogroup A: number analyzed (Participants) | 36 | 32
  Serogroup A | 13.7 [6.89 to 27.3] | 20.7 [9.96 to 43.2]
  Serogroup C: number analyzed (Participants) | 38 | 32
  Serogroup C | 251 [147 to 430] | 347 [230 to 523]
  Serogroup Y: number analyzed (Participants) | 36 | 25
  Serogroup Y | 152 [84.2 to 275] | 124 [56.3 to 276]
  Serogroup W: number analyzed (Participants) | 36 | 30
  Serogroup W | 87.1 [41.1 to 185] | 50.8 [19.4 to 133]

9. Secondary Outcome: Geometric Mean Titers of Antibodies Measured by rSBA Against Meningococcal Serogroups A, C, Y, and W Before Vaccination: Group 1 and 2 - PPAS3
Description: GMTs of antibody against meningococcal serogroups A, C, Y, and W were measured by rSBA. Titers were expressed in terms of 1/dilution.
Time Frame: Before vaccination at the age of 12 to 13 months
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 7 | 5
titers
  Serogroup A: number analyzed (Participants) | 6 | 5
  Serogroup A | 32.0 [1.20 to 855] | 169 [NA to NA] — 95% CI was not computable as the sample size was too small to compute valid data.
  Serogroup C | 58.0 [18.6 to 181] | 3.48 [NA to NA] — 95% CI was not computable as the sample size was too small to compute valid data.
  Serogroup Y | 58.0 [6.82 to 493] | 6.96 [NA to NA] — 95% CI was not computable as the sample size was too small to compute valid data.
  Serogroup W: number analyzed (Participants) | 5 | 5
  Serogroup W | 8.00 [NA to NA] — 95% CI was not computable as the sample size was too small to compute valid data. | 8.00 [NA to NA] — 95% CI was not computable as the sample size was too small to compute valid data.

10. Secondary Outcome: Geometric Mean Titers of Antibodies Measured by rSBA Against Meningococcal Serogroups A, C, Y, and W After Vaccination: Group 1 and 2 - PPAS3
Description: as for outcome 9
Time Frame: 30 days post-vaccination at the age of 12 to 13 months (i.e., at the age of 13 to 14 months)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 54 | 54
titers
  Serogroup A: number analyzed (Participants) | 47 | 43
  Serogroup A | 1741 [1354 to 2240] | 1508 [1073 to 2118]
  Serogroup C: number analyzed (Participants) | 47 | 43
  Serogroup C | 1396 [1047 to 1860] | 1532 [1061 to 2212]
  Serogroup Y: number analyzed (Participants) | 45 | 43
  Serogroup Y | 2620 [1999 to 3435] | 1414 [997 to 2005]
  Serogroup W: number analyzed (Participants) | 46 | 43
  Serogroup W | 2491 [1852 to 3351] | 2566 [1780 to 3700]

11. Secondary Outcome: Percentage of Participants With hSBA Antibody Titers >=1:4 and >=1:8 Against Meningococcal Serogroups A, C, Y, and W Before Vaccination: Group 1 and 2 - PPAS1
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by hSBA assay. Infancy was defined as up to 4 months of age. Percentage of participants with antibody titers >=1.4 and >=1:8 for meningococcal serogroups A, C, Y, and W were reported in this outcome measure.
Time Frame: Before vaccination at the age of 3 months
Population: Analysis was performed on PPAS1. Here, 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for Group 3.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 78 | 77
percentage of participants
  Serogroup A: >= 1:4: number analyzed (Participants) | 22 | 27
  Serogroup A: >= 1:4 | 81.8 [59.7 to 94.8] | 74.1 [53.7 to 88.9]
  Serogroup A: >= 1:8: number analyzed (Participants) | 22 | 27
  Serogroup A: >= 1:8 | 59.1 [36.4 to 79.3] | 48.1 [28.7 to 68.1]
  Serogroup C: >= 1:4: number analyzed (Participants) | 27 | 34
  Serogroup C: >= 1:4 | 55.6 [35.3 to 74.5] | 38.2 [22.2 to 56.4]
  Serogroup C: >= 1:8: number analyzed (Participants) | 27 | 34
  Serogroup C: >= 1:8 | 25.9 [11.1 to 46.3] | 20.6 [8.7 to 37.9]
  Serogroup Y: >= 1:4: number analyzed (Participants) | 27 | 30
  Serogroup Y: >= 1:4 | 29.6 [13.8 to 50.2] | 26.7 [12.3 to 45.9]
  Serogroup Y: >= 1:8: number analyzed (Participants) | 27 | 30
  Serogroup Y: >= 1:8 | 22.2 [8.6 to 42.3] | 10.0 [2.1 to 26.5]
  Serogroup W: >= 1:4: number analyzed (Participants) | 24 | 29
  Serogroup W: >= 1:4 | 16.7 [4.7 to 37.4] | 10.3 [2.2 to 27.4]
  Serogroup W: >= 1:8: number analyzed (Participants) | 24 | 29
  Serogroup W: >= 1:8 | 8.3 [1.0 to 27.0] | 0 [0 to 11.9]

12. Secondary Outcome: Percentage of Participants With hSBA Antibody Titers >=1:4 and >=1:8 Against Meningococcal Serogroups A, C, Y, and W After Vaccination: Group 1 and 2 - PPAS1
Description: as for outcome 11
Time Frame: 30 days post-vaccination at the age of 3 months (i.e., at the age of 4 months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 78 | 77
percentage of participants
  Serogroup A: >= 1:4: number analyzed (Participants) | 64 | 71
  Serogroup A: >= 1:4 | 87.5 [76.8 to 94.4] | 85.9 [75.6 to 93.0]
  Serogroup A: >= 1:8: number analyzed (Participants) | 64 | 71
  Serogroup A: >= 1:8 | 73.4 [60.9 to 83.7] | 66.2 [54.0 to 77.0]
  Serogroup C: >= 1:4: number analyzed (Participants) | 77 | 77
  Serogroup C: >= 1:4 | 93.5 [85.5 to 97.9] | 90.9 [82.2 to 96.3]
  Serogroup C: >= 1:8: number analyzed (Participants) | 77 | 77
  Serogroup C: >= 1:8 | 87.0 [77.4 to 93.6] | 88.3 [79.0 to 94.5]
  Serogroup Y: >= 1:4: number analyzed (Participants) | 71 | 68
  Serogroup Y: >= 1:4 | 81.7 [70.7 to 89.9] | 69.1 [56.7 to 79.8]
  Serogroup Y: >= 1:8: number analyzed (Participants) | 71 | 68
  Serogroup Y: >= 1:8 | 66.2 [54.0 to 77.0] | 54.4 [41.9 to 66.5]
  Serogroup W: >= 1:4: number analyzed (Participants) | 76 | 73
  Serogroup W: >= 1:4 | 56.6 [44.7 to 67.9] | 46.6 [34.8 to 58.6]
  Serogroup W: >= 1:8: number analyzed (Participants) | 76 | 73
  Serogroup W: >= 1:8 | 35.5 [24.9 to 47.3] | 27.4 [17.6 to 39.1]

13. Secondary Outcome: Percentage of Participants With hSBA Antibody Titers >=1:4 and >=1:8 Against Meningococcal Serogroups A, C, Y, and W Before Vaccination: Group 1 and 2 - PPAS3
Description: as for outcome 11
Time Frame: Before vaccination at the age of 12 to 13 months
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 35 | 26
percentage of participants
  Serogroup A: >= 1:4: number analyzed (Participants) | 31 | 26
  Serogroup A: >= 1:4 | 100 [88.8 to 100] | 96.2 [80.4 to 99.9]
  Serogroup A: >= 1:8: number analyzed (Participants) | 31 | 26
  Serogroup A: >= 1:8 | 93.5 [78.6 to 99.2] | 76.9 [56.4 to 91.0]
  Serogroup C: >= 1:4 | 94.3 [80.8 to 99.3] | 73.1 [52.2 to 88.4]
  Serogroup C: >= 1:8 | 85.7 [69.7 to 95.2] | 53.8 [33.4 to 73.4]
  Serogroup Y: >= 1:4: number analyzed (Participants) | 32 | 26
  Serogroup Y: >= 1:4 | 96.9 [83.8 to 99.9] | 88.5 [69.8 to 97.6]
  Serogroup Y: >= 1:8: number analyzed (Participants) | 32 | 26
  Serogroup Y: >= 1:8 | 93.8 [79.2 to 99.2] | 73.1 [52.2 to 88.4]
  Serogroup W: >= 1:4 | 97.1 [85.1 to 99.9] | 84.6 [65.1 to 95.6]
  Serogroup W: >= 1:8 | 88.6 [73.3 to 96.8] | 69.2 [48.2 to 85.7]

14. Secondary Outcome: Percentage of Participants With hSBA Antibody Titers >=1:4 and >=1:8 Against Meningococcal Serogroups A, C, Y, and W After Vaccination: Group 1 and 2 - PPAS3
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by hSBA assay. Percentage of participants with antibody titers >=1.4 and >=1:8 for meningococcal serogroups A, C, Y, and W were reported in this outcome measure.
Time Frame: 30 days post-vaccination at the age of 12 to 13 months (i.e., at the age of 13 to 14 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 178 | 169
percentage of participants
  Serogroup A: >= 1:4: number analyzed (Participants) | 159 | 156
  Serogroup A: >= 1:4 | 100 [97.7 to 100] | 100 [97.7 to 100]
  Serogroup A: >= 1:8: number analyzed (Participants) | 159 | 156
  Serogroup A: >= 1:8 | 100 [97.7 to 100] | 99.4 [96.5 to 100]
  Serogroup C: >= 1:4: number analyzed (Participants) | 168 | 165
  Serogroup C: >= 1:4 | 100 [97.8 to 100] | 100 [97.8 to 100]
  Serogroup C: >= 1:8: number analyzed (Participants) | 168 | 165
  Serogroup C: >= 1:8 | 100 [97.8 to 100] | 100 [97.8 to 100]
  Serogroup Y: >= 1:4: number analyzed (Participants) | 161 | 159
  Serogroup Y: >= 1:4 | 100 [97.7 to 100] | 100 [97.7 to 100]
  Serogroup Y: >= 1:8: number analyzed (Participants) | 161 | 159
  Serogroup Y: >= 1:8 | 100 [97.7 to 100] | 100 [97.7 to 100]
  Serogroup W: >= 1:4: number analyzed (Participants) | 172 | 160
  Serogroup W: >= 1:4 | 99.4 [96.8 to 100] | 100 [97.7 to 100]
  Serogroup W: >= 1:8: number analyzed (Participants) | 172 | 160
  Serogroup W: >= 1:8 | 99.4 [96.8 to 100] | 100 [97.7 to 100]

15. Secondary Outcome: Percentage of Participants With rSBA Antibody Titers >=1:8 and >=1:128 Against Meningococcal Serogroups A, C, Y, and W Before Vaccination: Group 1 and 2 - PPAS1
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by rSBA assay. Infancy was defined as up to 4 months of age. Percentage of participants with antibody titers >=1.8 and >=1:128 for meningococcal serogroups A, C, Y, and W were reported in this outcome measure.
Time Frame: Before vaccination at the age of 3 months
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 47 | 51
percentage of participants
  Serogroup A: >= 1:8: number analyzed (Participants) | 16 | 22
  Serogroup A: >= 1:8 | 0 [0 to 20.6] | 0 [0 to 15.4]
  Serogroup A: >= 1:128: number analyzed (Participants) | 16 | 22
  Serogroup A: >= 1:128 | 0 [0 to 20.6] | 0 [0 to 15.4]
  Serogroup C: >= 1:8: number analyzed (Participants) | 19 | 23
  Serogroup C: >= 1:8 | 15.8 [3.4 to 39.6] | 17.4 [5.0 to 38.8]
  Serogroup C: >= 1:128: number analyzed (Participants) | 19 | 23
  Serogroup C: >= 1:128 | 0 [0 to 17.6] | 4.3 [0.1 to 21.9]
  Serogroup Y: >= 1:8: number analyzed (Participants) | 19 | 23
  Serogroup Y: >= 1:8 | 10.5 [1.3 to 33.1] | 13.0 [2.8 to 33.6]
  Serogroup Y: >= 1:128: number analyzed (Participants) | 19 | 23
  Serogroup Y: >= 1:128 | 0 [0 to 17.6] | 0 [0 to 14.8]
  Serogroup W: >= 1:8: number analyzed (Participants) | 17 | 23
  Serogroup W: >= 1:8 | 11.8 [1.5 to 36.4] | 0 [0 to 14.8]
  Serogroup W: >= 1:128: number analyzed (Participants) | 17 | 23
  Serogroup W: >= 1:128 | 0 [0 to 19.5] | 0 [0 to 14.8]

16. Secondary Outcome: Percentage of Participants With rSBA Antibody Titers >=1:8 and >=1:128 Against Meningococcal Serogroups A, C, Y, and W After Vaccination: Group 1 and 2 - PPAS1
Description: as for outcome 15
Time Frame: 30 days post-vaccination at the age of 3 months (i.e., at the age of 4 months)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 47 | 51
percentage of participants
  Serogroup A: >= 1:8: number analyzed (Participants) | 36 | 32
  Serogroup A: >= 1:8 | 52.8 [35.5 to 69.6] | 65.6 [46.8 to 81.4]
  Serogroup A: >= 1:128: number analyzed (Participants) | 36 | 32
  Serogroup A: >= 1:128 | 19.4 [8.2 to 36.0] | 28.1 [13.7 to 46.7]
  Serogroup C: >= 1:8: number analyzed (Participants) | 38 | 32
  Serogroup C: >= 1:8 | 97.4 [86.2 to 99.9] | 100 [89.1 to 100]
  Serogroup C: >= 1:128: number analyzed (Participants) | 38 | 32
  Serogroup C: >= 1:128 | 78.9 [62.7 to 90.4] | 96.9 [83.8 to 99.9]
  Serogroup Y: >= 1:8: number analyzed (Participants) | 36 | 25
  Serogroup Y: >= 1:8 | 91.7 [77.5 to 98.2] | 92.0 [74.0 to 99.0]
  Serogroup Y: >= 1:128: number analyzed (Participants) | 36 | 25
  Serogroup Y: >= 1:128 | 80.6 [64.0 to 91.8] | 68.0 [46.5 to 85.1]
  Serogroup W: >= 1:8: number analyzed (Participants) | 36 | 30
  Serogroup W: >= 1:8 | 77.8 [60.8 to 89.9] | 63.3 [43.9 to 80.1]
  Serogroup W: >= 1:128: number analyzed (Participants) | 36 | 30
  Serogroup W: >= 1:128 | 75.0 [57.8 to 87.9] | 53.3 [34.3 to 71.7]

17. Secondary Outcome: Percentage of Participants With rSBA Antibody Titers >=1:8 and >=1:128 Against Meningococcal Serogroups A, C, Y, and W Before Vaccination: Group 1 and 2 - PPAS3
Description: as for outcome 15
Time Frame: Before vaccination at the age of 12 to 13 months
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 7 | 5
percentage of participants
  Serogroup A: >= 1:8: number analyzed (Participants) | 6 | 5
  Serogroup A: >= 1:8 | 50.0 [11.8 to 88.2] | 80.0 [28.4 to 99.5]
  Serogroup A: >= 1:128: number analyzed (Participants) | 6 | 5
  Serogroup A: >= 1:128 | 50.0 [11.8 to 88.2] | 80.0 [28.4 to 99.5]
  Serogroup C: >= 1:8 | 100 [59.0 to 100] | 20.0 [0.5 to 71.6]
  Serogroup C: >= 1:128 | 42.9 [9.9 to 81.6] | 0 [0 to 52.2]
  Serogroup Y: >= 1:8 | 85.7 [42.1 to 99.6] | 40.0 [5.3 to 85.3]
  Serogroup Y: >= 1:128 | 28.6 [3.7 to 71.0] | 0 [0 to 52.2]
  Serogroup W: >= 1:8: number analyzed (Participants) | 5 | 5
  Serogroup W: >= 1:8 | 40.0 [5.3 to 85.3] | 60.0 [14.7 to 94.7]
  Serogroup W: >= 1:128: number analyzed (Participants) | 5 | 5
  Serogroup W: >= 1:128 | 20.0 [0.5 to 71.6] | 0 [0 to 52.2]

18. Secondary Outcome: Percentage of Participants With rSBA Antibody Titers >=1:8 and >=1:128 Against Meningococcal Serogroups A, C, Y, and W After Vaccination: Group 1 and 2 - PPAS3
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by rSBA assay. Percentage of participants with antibody titers >=1.8 and >=1:128 for meningococcal serogroups A, C, Y, and W were reported in this outcome measure.
Time Frame: 30 days post-vaccination at the age of 12 to 13 months (i.e., at the age of 13 to 14 months)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 54 | 54
percentage of participants
  Serogroup A: >= 1:8: number analyzed (Participants) | 47 | 43
  Serogroup A: >= 1:8 | 100 [92.5 to 100] | 100 [91.8 to 100]
  Serogroup A: >= 1:128: number analyzed (Participants) | 47 | 43
  Serogroup A: >= 1:128 | 100 [92.5 to 100] | 97.7 [87.7 to 99.9]
  Serogroup C: >= 1:8: number analyzed (Participants) | 47 | 43
  Serogroup C: >= 1:8 | 100 [92.5 to 100] | 100 [91.8 to 100]
  Serogroup C: >= 1:128: number analyzed (Participants) | 47 | 43
  Serogroup C: >= 1:128 | 100 [92.5 to 100] | 100 [91.8 to 100]
  Serogroup Y: >= 1:8: number analyzed (Participants) | 45 | 43
  Serogroup Y: >= 1:8 | 100 [92.1 to 100] | 100 [91.8 to 100]
  Serogroup Y: >= 1:128: number analyzed (Participants) | 45 | 43
  Serogroup Y: >= 1:128 | 100 [92.1 to 100] | 97.7 [87.7 to 99.9]
  Serogroup W: >= 1:8: number analyzed (Participants) | 46 | 43
  Serogroup W: >= 1:8 | 100 [92.3 to 100] | 100 [91.8 to 100]
  Serogroup W: >= 1:128: number analyzed (Participants) | 46 | 43
  Serogroup W: >= 1:128 | 100 [92.3 to 100] | 97.7 [87.7 to 99.9]

19. Secondary Outcome: Percentage of Participants With >= 4-Fold Rise in hSBA Antibody Titers Against Meningococcal Serogroups A, C, Y, and W After Vaccination: Group 1 and 2 - PPAS1
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by hSBA assay. Fold-rise was calculated as ratio of post-vaccination titer (i.e., 30 days post-vaccination at the age of 3 months) to pre-dose titer at the age of 3 months. Infancy was defined as up to 4 months of age.
Time Frame: Before vaccination at the age of 3 months, 30 days post-vaccination at the age of 3 months (i.e., at the age of 4 months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 78 | 77
percentage of participants
  Serogroup A: number analyzed (Participants) | 17 | 24
  Serogroup A | 5.9 [0.1 to 28.7] | 25.0 [9.8 to 46.7]
  Serogroup C: number analyzed (Participants) | 27 | 34
  Serogroup C | 70.4 [49.8 to 86.2] | 82.4 [65.5 to 93.2]
  Serogroup Y: number analyzed (Participants) | 24 | 26
  Serogroup Y | 45.8 [25.6 to 67.2] | 53.8 [33.4 to 73.4]
  Serogroup W: number analyzed (Participants) | 24 | 27
  Serogroup W | 29.2 [12.6 to 51.1] | 18.5 [6.3 to 38.1]

20. Secondary Outcome: Percentage of Participants With >= 4-Fold Rise in hSBA Antibody Titers Against Meningococcal Serogroups A, C, Y, and W After Vaccination: Group 1 and 2 - PPAS3
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by hSBA assay. Fold-rise was calculated as ratio of post-vaccination titer (i.e., 30 days post-vaccination at the age of 12 to 13 months) to pre-dose titer before vaccination at the age of 3 months.
Time Frame: Before vaccination at the age of 3 months, 30 days post-vaccination at the age of 12 to 13 months (i.e., at the age of 13 to 14 months)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 28 | 32
percentage of participants
  Serogroup A: number analyzed (Participants) | 22 | 24
  Serogroup A | 100 [84.6 to 100] | 91.7 [73.0 to 99.0]
  Serogroup C | 92.9 [76.5 to 99.1] | 93.8 [79.2 to 99.2]
  Serogroup Y: number analyzed (Participants) | 27 | 29
  Serogroup Y | 96.3 [81.0 to 99.9] | 100 [88.1 to 100]
  Serogroup W: number analyzed (Participants) | 26 | 26
  Serogroup W | 100 [86.8 to 100] | 100 [86.8 to 100]

21. Secondary Outcome: Percentage of Participants With >= 4-Fold Rise in hSBA Antibody Titers Against Meningococcal Serogroups A, C, Y, and W After Vaccination: Group 1 and 2 - PPAS3
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by hSBA assay. Fold-rise was calculated as ratio of post-vaccination titer (i.e., 30 days post-vaccination at the age of 12 to 13 months) to pre-dose titer before vaccination at the age of 12 to 13 months.
Time Frame: Before vaccination at the age of 12 to 13 months, 30 days post-vaccination at the age of 12 to 13 months (i.e., at the age of 13 to 14 months)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 34 | 26
percentage of participants
  Serogroup A: number analyzed (Participants) | 27 | 26
  Serogroup A | 100 [87.2 to 100] | 53.8 [33.4 to 73.4]
  Serogroup C: number analyzed (Participants) | 33 | 26
  Serogroup C | 100 [89.4 to 100] | 100 [86.8 to 100]
  Serogroup Y: number analyzed (Participants) | 29 | 25
  Serogroup Y | 89.7 [72.6 to 97.8] | 96.0 [79.6 to 99.9]
  Serogroup W: number analyzed (Participants) | 34 | 25
  Serogroup W | 85.3 [68.9 to 95.0] | 100 [86.3 to 100]

22. Secondary Outcome: Percentage of Participants With >= 4-Fold Rise in rSBA Antibody Titers Against Meningococcal Serogroups A, C, Y, and W After Vaccination: Group 1 and 2 - PPAS1
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by rSBA assay. Fold-rise was calculated as ratio of post-vaccination titer (i.e., 30 days post-vaccination at the age of 3 months) to pre-dose titer at the age of 3 months. Infancy was defined as up to 4 months of age.
Time Frame: as for outcome 19
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 47 | 51
percentage of participants
  Serogroup A: number analyzed (Participants) | 13 | 16
  Serogroup A | 46.2 [19.2 to 74.9] | 62.5 [35.4 to 84.8]
  Serogroup C: number analyzed (Participants) | 15 | 16
  Serogroup C | 86.7 [59.5 to 98.3] | 87.5 [61.7 to 98.4]
  Serogroup Y: number analyzed (Participants) | 14 | 11
  Serogroup Y | 78.6 [49.2 to 95.3] | 90.9 [58.7 to 99.8]
  Serogroup W: number analyzed (Participants) | 14 | 15
  Serogroup W | 57.1 [28.9 to 82.3] | 53.3 [26.6 to 78.7]

23. Secondary Outcome: Percentage of Participants With >= 4-Fold Rise in rSBA Antibody Titers Against Meningococcal Serogroups A, C, Y, and W After Vaccination: Group 1 and 2 - PPAS3
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by rSBA assay. Fold-rise was calculated as ratio of post-vaccination titer (i.e., 30 days post-vaccination at the age of 12 to 13 months) to pre-dose titer before vaccination at the age of 3 months.
Time Frame: as for outcome 20
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 54 | 54
percentage of participants
  Serogroup A: number analyzed (Participants) | 13 | 17
  Serogroup A | 100 [75.3 to 100] | 100 [80.5 to 100]
  Serogroup C: number analyzed (Participants) | 17 | 17
  Serogroup C | 100 [80.5 to 100] | 100 [80.5 to 100]
  Serogroup Y: number analyzed (Participants) | 16 | 17
  Serogroup Y | 100 [79.4 to 100] | 100 [80.5 to 100]
  Serogroup W: number analyzed (Participants) | 15 | 17
  Serogroup W | 100 [78.2 to 100] | 100 [80.5 to 100]

24. Secondary Outcome: Percentage of Participants With >= 4-Fold Rise in rSBA Antibody Titers Against Meningococcal Serogroups A, C, Y, and W After Vaccination: Group 1 and 2 - PPAS3
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by rSBA assay. Fold-rise was calculated as ratio of post-vaccination titer (i.e., 30 days post-vaccination at the age of 12 to 13 months) to pre-dose titer before vaccination at the age of 12 to 13 months.
Time Frame: as for outcome 21
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 7 | 5
percentage of participants
  Serogroup A: number analyzed (Participants) | 6 | 5
  Serogroup A | 83.3 [35.9 to 99.6] | 100 [47.8 to 100]
  Serogroup C | 100 [59.0 to 100] | 100 [47.8 to 100]
  Serogroup Y | 71.4 [29.0 to 96.3] | 100 [47.8 to 100]
  Serogroup W: number analyzed (Participants) | 5 | 5
  Serogroup W | 100 [47.8 to 100] | 100 [47.8 to 100]

25. Secondary Outcome: Percentage of Participants With Vaccine Seroresponse Measured by hSBA Against Meningococcal Serogroups A, C, Y, and W After Vaccination: Group 1 and 2 - PPAS1
Description: The hSBA vaccine seroresponse against serogroups A, C, Y, and W was defined as post-vaccination hSBA titer >=1:16 for participants with pre-vaccination hSBA titer <1:8 or at least a 4-fold increase in hSBA titers from pre to post-vaccination for participants with pre-vaccination hSBA titers >=1:8. Infancy was defined as up to 4 months of age.
Time Frame: Before vaccination at the age of 3 months up to 30 days post-vaccination at the age of 3 months (i.e., at the age of 4 months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 78 | 77
percentage of participants
  Serogroup A: number analyzed (Participants) | 17 | 24
  Serogroup A | 0 [0 to 19.5] | 20.8 [7.1 to 42.2]
  Serogroup C: number analyzed (Participants) | 27 | 34
  Serogroup C | 66.7 [46.0 to 83.5] | 79.4 [62.1 to 91.3]
  Serogroup Y: number analyzed (Participants) | 24 | 26
  Serogroup Y | 33.3 [15.6 to 55.3] | 30.8 [14.3 to 51.8]
  Serogroup W: number analyzed (Participants) | 24 | 27
  Serogroup W | 25.0 [9.8 to 46.7] | 11.1 [2.4 to 29.2]

26. Secondary Outcome: Percentage of Participants With Vaccine Seroresponse Measured by hSBA Against Meningococcal Serogroups A, C, Y, and W After Vaccination: Group 1 and 2 - PPAS3
Description: The hSBA vaccine seroresponse against serogroups A, C, Y, and W was defined as post-vaccination hSBA titer >=1:16 for participants with pre-vaccination hSBA titer <1:8 or at least a 4-fold increase in hSBA titers from pre to post-vaccination for participants with pre-vaccination hSBA titers >=1:8.
Time Frame: Before vaccination at the age of 3 months up to 30 days post-vaccination at the age of 12 to 13 months (i.e., at the age of 13 to 14 months)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 28 | 32
percentage of participants
  Serogroup A: number analyzed (Participants) | 22 | 24
  Serogroup A | 100 [84.6 to 100] | 91.7 [73.0 to 99.0]
  Serogroup C | 92.9 [76.5 to 99.1] | 93.8 [79.2 to 99.2]
  Serogroup Y: number analyzed (Participants) | 27 | 29
  Serogroup Y | 96.3 [81.0 to 99.9] | 96.6 [82.2 to 99.9]
  Serogroup W: number analyzed (Participants) | 26 | 26
  Serogroup W | 100 [86.8 to 100] | 100 [86.8 to 100]

27. Secondary Outcome: Percentage of Participants With Vaccine Seroresponse Measured by hSBA Against Meningococcal Serogroups A, C, Y, and W After Vaccination: Group 1 and 2 - PPAS3
Description: as for outcome 26
Time Frame: Before vaccination at the age of 12 to 13 months up to 30 days post-vaccination at the age of 12 to 13 months (i.e., at the age of 13 to 14 months)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 34 | 26
percentage of participants
  Serogroup A: number analyzed (Participants) | 27 | 26
  Serogroup A | 100 [87.2 to 100] | 53.8 [33.4 to 73.4]
  Serogroup C: number analyzed (Participants) | 33 | 26
  Serogroup C | 100 [89.4 to 100] | 96.2 [80.4 to 99.9]
  Serogroup Y: number analyzed (Participants) | 29 | 25
  Serogroup Y | 89.7 [72.6 to 97.8] | 96.0 [79.6 to 99.9]
  Serogroup W: number analyzed (Participants) | 34 | 25
  Serogroup W | 85.3 [68.9 to 95.0] | 100 [86.3 to 100]

28. Secondary Outcome: Percentage of Participants With Vaccine Seroresponse Measured by rSBA Against Meningococcal Serogroups A, C, Y, and W After Vaccination: Group 1 and 2 - PPAS1
Description: The rSBA vaccine seroresponse against serogroups A, C, Y, and W was defined as post-vaccination rSBA titer >=1:32 for participants with pre-vaccination rSBA titer <1:8 or at least a 4-fold increase in hSBA titers from pre to post-vaccination for participants with pre-vaccination hSBA titers >=1:8. Infancy was defined as up to 4 months of age.
Time Frame: as for outcome 25
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 47 | 51
percentage of participants
  Serogroup A: number analyzed (Participants) | 13 | 16
  Serogroup A | 30.8 [9.1 to 61.4] | 50.0 [24.7 to 75.3]
  Serogroup C: number analyzed (Participants) | 15 | 16
  Serogroup C | 86.7 [59.5 to 98.3] | 87.5 [61.7 to 98.4]
  Serogroup Y: number analyzed (Participants) | 14 | 11
  Serogroup Y | 71.4 [41.9 to 91.6] | 72.7 [39.0 to 94.0]
  Serogroup W: number analyzed (Participants) | 14 | 15
  Serogroup W | 57.1 [28.9 to 82.3] | 53.3 [26.6 to 78.7]

29. Secondary Outcome: Percentage of Participants With Vaccine Seroresponse Measured by rSBA Against Meningococcal Serogroups A, C, Y, and W After Vaccination: Group 1 and 2 - PPAS3
Description: The rSBA vaccine seroresponse against serogroups A, C, Y, and W was defined as post-vaccination rSBA titer >=1:32 for participants with pre-vaccination rSBA titer <1:8 or at least a 4-fold increase in hSBA titers from pre to post-vaccination for participants with pre-vaccination hSBA titers >=1:8.
Time Frame: as for outcome 26
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 54 | 54
percentage of participants
  Serogroup A: number analyzed (Participants) | 13 | 17
  Serogroup A | 100 [75.3 to 100] | 100 [80.5 to 100]
  Serogroup C: number analyzed (Participants) | 17 | 17
  Serogroup C | 100 [80.5 to 100] | 100 [80.5 to 100]
  Serogroup Y: number analyzed (Participants) | 16 | 17
  Serogroup Y | 100 [79.4 to 100] | 94.1 [71.3 to 99.9]
  Serogroup W: number analyzed (Participants) | 15 | 17
  Serogroup W | 100 [78.2 to 100] | 100 [80.5 to 100]

30. Secondary Outcome: Percentage of Participants With Vaccine Seroresponse Measured by rSBA Against Meningococcal Serogroups A, C, Y, and W After Vaccination: Group 1 and 2 - PPAS3
Description: as for outcome 29
Time Frame: as for outcome 27
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 7 | 5
percentage of participants
  Serogroup A: number analyzed (Participants) | 6 | 5
  Serogroup A | 83.3 [35.9 to 99.6] | 100 [47.8 to 100]
  Serogroup C | 100 [59.0 to 100] | 100 [47.8 to 100]
  Serogroup Y | 71.4 [29.0 to 96.3] | 100 [47.8 to 100]
  Serogroup W: number analyzed (Participants) | 5 | 5
  Serogroup W | 100 [47.8 to 100] | 100 [47.8 to 100]

31. Secondary Outcome: Percentage of Participants With Distribution of hSBA Titers Against Meningococcal Serogroups A, C, Y, and W Before Vaccination - PPAS1
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by hSBA assay. Percentage of participants with hSBA antibody titers distribution <1:4, >=1:4, >=1:8, >=1:16; >=1:32; >=1:64, >=1:128, >=1:256; >=1:512; >=1:1024 for meningococcal serogroups A, C, Y, and W were reported in this outcome measure.
Time Frame: Before vaccination at the age of 3 months
Population: Analysis was performed on PPAS1. Here, 'number analyzed' = participants with available data for each specified category and '0' in the number analyzed field denotes that no participant had available data for the specified titer category.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months) | Group 3: Bexsero® (2, 4, and 12 to 13 Months)
Number analyzed (Participants) | 78 | 77 | 84
percentage of participants
  Serogroup A: <1:4: number analyzed (Participants) | 22 | 27 | 29
  Serogroup A: <1:4 | 18.2 | 25.9 | 24.1
  Serogroup A: >=1:4: number analyzed (Participants) | 22 | 27 | 29
  Serogroup A: >=1:4 | 81.8 | 74.1 | 75.9
  Serogroup A: >=1:8: number analyzed (Participants) | 22 | 27 | 29
  Serogroup A: >=1:8 | 59.1 | 48.1 | 48.3
  Serogroup A: >=1:16: number analyzed (Participants) | 22 | 27 | 29
  Serogroup A: >=1:16 | 36.4 | 33.3 | 27.6
  Serogroup A: >=1:32: number analyzed (Participants) | 22 | 27 | 29
  Serogroup A: >=1:32 | 22.7 | 11.1 | 20.7
  Serogroup A: >=1:64: number analyzed (Participants) | 22 | 27 | 29
  Serogroup A: >=1:64 | 4.5 | 7.4 | 10.3
  Serogroup A: >=1:128: number analyzed (Participants) | 22 | 27 | 29
  Serogroup A: >=1:128 | 4.5 | 7.4 | 3.4
  Serogroup A: >=1:256: number analyzed (Participants) | 22 | 27 | 0
  Serogroup A: >=1:256 | 0 | 3.7 |
  Serogroup A: >=1:512: number analyzed (Participants) | 22 | 27 | 0
  Serogroup A: >=1:512 | 0 | 0 |
  Serogroup A: >=1:1024: number analyzed (Participants) | 22 | 27 | 0
  Serogroup A: >=1:1024 | 0 | 0 |
  Serogroup C: <1:4: number analyzed (Participants) | 27 | 34 | 35
  Serogroup C: <1:4 | 44.4 | 61.8 | 62.9
  Serogroup C: >=1:4: number analyzed (Participants) | 27 | 34 | 35
  Serogroup C: >=1:4 | 55.6 | 38.2 | 37.1
  Serogroup C: >=1:8: number analyzed (Participants) | 27 | 34 | 35
  Serogroup C: >=1:8 | 25.9 | 20.6 | 14.3
  Serogroup C: >=1:16: number analyzed (Participants) | 27 | 34 | 35
  Serogroup C: >=1:16 | 7.4 | 11.8 | 11.4
  Serogroup C: >=1:32: number analyzed (Participants) | 27 | 34 | 35
  Serogroup C: >=1:32 | 0 | 5.9 | 2.9
  Serogroup C: >=1:64: number analyzed (Participants) | 27 | 34 | 35
  Serogroup C: >=1:64 | 0 | 5.9 | 2.9
  Serogroup C: >=1:128: number analyzed (Participants) | 27 | 34 | 35
  Serogroup C: >=1:128 | 0 | 5.9 | 0
  Serogroup C: >=1:256: number analyzed (Participants) | 27 | 34 | 0
  Serogroup C: >=1:256 | 0 | 2.9 |
  Serogroup C: >=1:512: number analyzed (Participants) | 27 | 34 | 0
  Serogroup C: >=1:512 | 0 | 2.9 |
  Serogroup C: >=1:1024: number analyzed (Participants) | 27 | 34 | 0
  Serogroup C: >=1:1024 | 0 | 0 |
  Serogroup Y: <1:4: number analyzed (Participants) | 27 | 30 | 33
  Serogroup Y: <1:4 | 70.4 | 73.3 | 84.8
  Serogroup Y: >=1:4: number analyzed (Participants) | 27 | 30 | 33
  Serogroup Y: >=1:4 | 29.6 | 26.7 | 15.2
  Serogroup Y: >=1:8: number analyzed (Participants) | 27 | 30 | 33
  Serogroup Y: >=1:8 | 22.2 | 10.0 | 12.1
  Serogroup Y: >=1:16: number analyzed (Participants) | 27 | 30 | 33
  Serogroup Y: >=1:16 | 7.4 | 0 | 3.0
  Serogroup Y: >=1:32: number analyzed (Participants) | 27 | 30 | 33
  Serogroup Y: >=1:32 | 3.7 | 0 | 0
  Serogroup Y: >=1:64: number analyzed (Participants) | 27 | 30 | 33
  Serogroup Y: >=1:64 | 3.7 | 0 | 0
  Serogroup Y: >=1:128: number analyzed (Participants) | 27 | 30 | 33
  Serogroup Y: >=1:128 | 3.7 | 0 | 0
  Serogroup Y: >=1:256: number analyzed (Participants) | 27 | 30 | 0
  Serogroup Y: >=1:256 | 0 | 0 |
  Serogroup Y: >=1:512: number analyzed (Participants) | 27 | 30 | 0
  Serogroup Y: >=1:512 | 0 | 0 |
  Serogroup Y: >=1:1024: number analyzed (Participants) | 27 | 30 | 0
  Serogroup Y: >=1:1024 | 0 | 0 |
  Serogroup W: <1:4: number analyzed (Participants) | 24 | 29 | 32
  Serogroup W: <1:4 | 83.3 | 89.7 | 87.5
  Serogroup W: >=1:4: number analyzed (Participants) | 24 | 29 | 32
  Serogroup W: >=1:4 | 16.7 | 10.3 | 12.5
  Serogroup W: >=1:8: number analyzed (Participants) | 24 | 29 | 32
  Serogroup W: >=1:8 | 8.3 | 0 | 3.1
  Serogroup W: >=1:16: number analyzed (Participants) | 24 | 29 | 32
  Serogroup W: >=1:16 | 4.2 | 0 | 3.1
  Serogroup W: >=1:32: number analyzed (Participants) | 24 | 29 | 32
  Serogroup W: >=1:32 | 4.2 | 0 | 3.1
  Serogroup W: >=1:64: number analyzed (Participants) | 24 | 29 | 32
  Serogroup W: >=1:64 | 0 | 0 | 0
  Serogroup W: >=1:128: number analyzed (Participants) | 24 | 29 | 32
  Serogroup W: >=1:128 | 0 | 0 | 0
  Serogroup W: >=1:256: number analyzed (Participants) | 24 | 29 | 0
  Serogroup W: >=1:256 | 0 | 0 |
  Serogroup W: >=1:512: number analyzed (Participants) | 24 | 29 | 0
  Serogroup W: >=1:512 | 0 | 0 |
  Serogroup W: >=1:1024: number analyzed (Participants) | 24 | 29 | 0
  Serogroup W: >=1:1024 | 0 | 0 |

32. Secondary Outcome: Percentage of Participants With Distribution of hSBA Titers Against Meningococcal Serogroups A, C, Y, and W After Vaccination - PPAS1
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by hSBA assay. Infancy was defined as up to 4 months of age. Percentage of participants with hSBA antibody titers distribution <1:4, >=1:4, >=1:8, >=1:16; >=1:32; >=1:64, >=1:128, >=1:256; >=1:512; >=1:1024 for meningococcal serogroups A, C, Y, and W were reported in this outcome measure.
Time Frame: 30 days post-vaccination at the age of 3 months (i.e., at the age of 4 months)
Population: as for outcome 31
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months) | Group 3: Bexsero® (2, 4, and 12 to 13 Months)
Number analyzed (Participants) | 78 | 77 | 84
percentage of participants
  Serogroup A: <1:4: number analyzed (Participants) | 64 | 71 | 66
  Serogroup A: <1:4 | 12.5 | 14.1 | 21.2
  Serogroup A: >=1:4: number analyzed (Participants) | 64 | 71 | 66
  Serogroup A: >=1:4 | 87.5 | 85.9 | 78.8
  Serogroup A: >=1:8: number analyzed (Participants) | 64 | 71 | 66
  Serogroup A: >=1:8 | 73.4 | 66.2 | 51.5
  Serogroup A: >=1:16: number analyzed (Participants) | 64 | 71 | 66
  Serogroup A: >=1:16 | 51.6 | 42.3 | 34.8
  Serogroup A: >=1:32: number analyzed (Participants) | 64 | 71 | 66
  Serogroup A: >=1:32 | 21.9 | 19.7 | 16.7
  Serogroup A: >=1:64: number analyzed (Participants) | 64 | 71 | 66
  Serogroup A: >=1:64 | 7.8 | 9.9 | 9.1
  Serogroup A: >=1:128: number analyzed (Participants) | 64 | 71 | 66
  Serogroup A: >=1:128 | 1.6 | 2.8 | 3.0
  Serogroup A: >=1:256: number analyzed (Participants) | 64 | 71 | 0
  Serogroup A: >=1:256 | 0 | 0 |
  Serogroup A: >=1:512: number analyzed (Participants) | 64 | 71 | 0
  Serogroup A: >=1:512 | 0 | 0 |
  Serogroup A: >=1:1024: number analyzed (Participants) | 64 | 71 | 0
  Serogroup A: >=1:1024 | 0 | 0 |
  Serogroup C: <1:4: number analyzed (Participants) | 77 | 77 | 84
  Serogroup C: <1:4 | 6.5 | 9.1 | 78.6
  Serogroup C: >=1:4: number analyzed (Participants) | 77 | 77 | 84
  Serogroup C: >=1:4 | 93.5 | 90.9 | 21.4
  Serogroup C: >=1:8: number analyzed (Participants) | 77 | 77 | 84
  Serogroup C: >=1:8 | 87.0 | 88.3 | 7.1
  Serogroup C: >=1:16: number analyzed (Participants) | 77 | 77 | 84
  Serogroup C: >=1:16 | 85.7 | 80.5 | 6.0
  Serogroup C: >=1:32: number analyzed (Participants) | 77 | 77 | 84
  Serogroup C: >=1:32 | 81.8 | 71.4 | 3.6
  Serogroup C: >=1:64: number analyzed (Participants) | 77 | 77 | 84
  Serogroup C: >=1:64 | 66.2 | 66.2 | 1.2
  Serogroup C: >=1:128: number analyzed (Participants) | 77 | 77 | 84
  Serogroup C: >=1:128 | 54.5 | 49.4 | 0
  Serogroup C: >=1:256: number analyzed (Participants) | 77 | 77 | 0
  Serogroup C: >=1:256 | 32.5 | 28.6 |
  Serogroup C: >=1:512: number analyzed (Participants) | 77 | 77 | 0
  Serogroup C: >=1:512 | 20.8 | 13.0 |
  Serogroup C: >=1:1024: number analyzed (Participants) | 77 | 77 | 0
  Serogroup C: >=1:1024 | 6.5 | 5.2 |
  Serogroup Y: <1:4: number analyzed (Participants) | 71 | 68 | 73
  Serogroup Y: <1:4 | 18.3 | 30.9 | 89.0
  Serogroup Y: >=1:4: number analyzed (Participants) | 71 | 68 | 73
  Serogroup Y: >=1:4 | 81.7 | 69.1 | 11.0
  Serogroup Y: >=1:8: number analyzed (Participants) | 71 | 68 | 73
  Serogroup Y: >=1:8 | 66.2 | 54.4 | 2.7
  Serogroup Y: >=1:16: number analyzed (Participants) | 71 | 68 | 73
  Serogroup Y: >=1:16 | 40.8 | 25.0 | 2.7
  Serogroup Y: >=1:32: number analyzed (Participants) | 71 | 68 | 73
  Serogroup Y: >=1:32 | 21.1 | 11.8 | 1.4
  Serogroup Y: >=1:64: number analyzed (Participants) | 71 | 68 | 73
  Serogroup Y: >=1:64 | 7.0 | 4.4 | 1.4
  Serogroup Y: >=1:128: number analyzed (Participants) | 71 | 68 | 73
  Serogroup Y: >=1:128 | 4.2 | 1.5 | 0
  Serogroup Y: >=1:256: number analyzed (Participants) | 71 | 68 | 0
  Serogroup Y: >=1:256 | 1.4 | 0 |
  Serogroup Y: >=1:512: number analyzed (Participants) | 71 | 68 | 0
  Serogroup Y: >=1:512 | 1.4 | 0 |
  Serogroup Y: >=1:1024: number analyzed (Participants) | 71 | 68 | 0
  Serogroup Y: >=1:1024 | 0 | 0 |
  Serogroup W: <1:4: number analyzed (Participants) | 76 | 73 | 77
  Serogroup W: <1:4 | 43.4 | 53.4 | 94.8
  Serogroup W: >=1:4: number analyzed (Participants) | 76 | 73 | 77
  Serogroup W: >=1:4 | 56.6 | 46.6 | 5.2
  Serogroup W: >=1:8: number analyzed (Participants) | 76 | 73 | 77
  Serogroup W: >=1:8 | 35.5 | 27.4 | 2.6
  Serogroup W: >=1:16: number analyzed (Participants) | 76 | 73 | 77
  Serogroup W: >=1:16 | 21.1 | 13.7 | 1.3
  Serogroup W: >=1:32: number analyzed (Participants) | 76 | 73 | 77
  Serogroup W: >=1:32 | 5.3 | 4.1 | 0
  Serogroup W: >=1:64: number analyzed (Participants) | 76 | 73 | 77
  Serogroup W: >=1:64 | 2.6 | 1.4 | 0
  Serogroup W: >=1:128: number analyzed (Participants) | 76 | 73 | 77
  Serogroup W: >=1:128 | 1.3 | 0 | 0
  Serogroup W: >=1:256: number analyzed (Participants) | 76 | 73 | 0
  Serogroup W: >=1:256 | 0 | 0 |
  Serogroup W: >=1:512: number analyzed (Participants) | 76 | 73 | 0
  Serogroup W: >=1:512 | 0 | 0 |
  Serogroup W: >=1:1024: number analyzed (Participants) | 76 | 73 | 0
  Serogroup W: >=1:1024 | 0 | 0 |

33. Secondary Outcome: Percentage of Participants With Distribution of hSBA Titers Against Meningococcal Serogroups A, C, Y, and W Before Vaccination - PPAS3
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by hSBA assay. Infancy was defined as up to 4 months of age. Percentage of participants with hSBA antibody titers distribution <1:4, >=1:4, >=1:8, >=1:16; >=1:32; >=1:64, >=1:128, >=1:256; >=1:512; >=1:1024; >=1:2048; >=1:4096; >=1:8192; >=1:16384; >=1:32768; >=1:65536 for meningococcal serogroups A, C, Y, and W were reported in this outcome measure.
Time Frame: Before vaccination at the age of 12 to 13 months
Population: Analysis was performed on PPAS3. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified category. Here, '0' in the number analyzed field denotes that no participant had available data for the specified titer category.
Measure: Number; unit: percentage of participants
Groups:
- Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months): Participants aged 2 months (at the time of enrollment) received MenACYW conjugate vaccine at 3 months and at 12 to 13 months of age, Bexsero® at 2, 4, and 12 to 13 months of age concomitantly with routine pediatric vaccines: Infanrix hexa® vaccine at 2, 3, and 4 months of age; Rotarix® vaccine at 2 and 3 months of age; Prevenar 13® vaccine at 2 and 4 months of age.
- Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months): Participants aged 2 months (at the time of enrollment) received MenACYW conjugate vaccine at 3 months and at 12 to 13 months of age, Bexsero® at 2 and 4 months of age concomitantly with routine pediatric vaccines: Infanrix hexa® vaccine at 2, 3, and 4 months of age; Rotarix® vaccine at 2 and 3 months of age; Prevenar 13® vaccine at 2 and 4 months of age.
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months) | Group 3: Bexsero® (2, 4, and 12 to 13 Months)
Number analyzed (Participants) | 35 | 26 | 35
percentage of participants
  Serogroup A: <1:4: number analyzed (Participants) | 31 | 26 | 34
  Serogroup A: <1:4 | 0 | 3.8 | 11.8
  Serogroup A: >=1:4: number analyzed (Participants) | 31 | 26 | 34
  Serogroup A: >=1:4 | 100 | 96.2 | 88.2
  Serogroup A: >=1:8: number analyzed (Participants) | 31 | 26 | 34
  Serogroup A: >=1:8 | 93.5 | 76.9 | 73.5
  Serogroup A: >=1:16: number analyzed (Participants) | 31 | 26 | 34
  Serogroup A: >=1:16 | 90.3 | 73.1 | 55.9
  Serogroup A: >=1:32: number analyzed (Participants) | 31 | 26 | 34
  Serogroup A: >=1:32 | 64.5 | 61.5 | 41.2
  Serogroup A: >=1:64: number analyzed (Participants) | 31 | 26 | 34
  Serogroup A: >=1:64 | 48.4 | 23.1 | 29.4
  Serogroup A: >=1:128: number analyzed (Participants) | 31 | 26 | 34
  Serogroup A: >=1:128 | 29.0 | 15.4 | 23.5
  Serogroup A: >=1:256: number analyzed (Participants) | 31 | 26 | 34
  Serogroup A: >=1:256 | 22.6 | 3.8 | 5.9
  Serogroup A: >=1:512: number analyzed (Participants) | 31 | 26 | 34
  Serogroup A: >=1:512 | 3.2 | 0 | 2.9
  Serogroup A: >=1:1024: number analyzed (Participants) | 31 | 26 | 34
  Serogroup A: >=1:1024 | 0 | 0 | 0
  Serogroup A: >=1:2048: number analyzed (Participants) | 31 | 26 | 34
  Serogroup A: >=1:2048 | 0 | 0 | 0
  Serogroup A: >=1:4096: number analyzed (Participants) | 31 | 26 | 34
  Serogroup A: >=1:4096 | 0 | 0 | 0
  Serogroup A: >=1:8192: number analyzed (Participants) | 31 | 26 | 34
  Serogroup A: >=1:8192 | 0 | 0 | 0
  Serogroup A: >=1:16384: number analyzed (Participants) | 31 | 26 | 34
  Serogroup A: >=1:16384 | 0 | 0 | 0
  Serogroup A: >=1:32768: number analyzed (Participants) | 31 | 26 | 34
  Serogroup A: >=1:32768 | 0 | 0 | 0
  Serogroup A: >=1:65536: number analyzed (Participants) | 0 | 0 | 34
  Serogroup A: >=1:65536 |  |  | 0
  Serogroup C: <1:4 | 5.7 | 26.9 | 94.3
  Serogroup C: >=1:4 | 94.3 | 73.1 | 5.7
  Serogroup C: >=1:8 | 85.7 | 53.8 | 0
  Serogroup C: >=1:16 | 71.4 | 42.3 | 0
  Serogroup C: >=1:32 | 65.7 | 34.6 | 0
  Serogroup C: >=1:64 | 48.6 | 3.8 | 0
  Serogroup C: >=1:128 | 20.0 | 0 | 0
  Serogroup C: >=1:256 | 5.7 | 0 | 0
  Serogroup C: >=1:512 | 0 | 0 | 0
  Serogroup C: >=1:1024 | 0 | 0 | 0
  Serogroup C: >=1:2048 | 0 | 0 | 0
  Serogroup C: >=1:4096 | 0 | 0 | 0
  Serogroup C: >=1:8192 | 0 | 0 | 0
  Serogroup C: >=1:16384 | 0 | 0 | 0
  Serogroup C: >=1:32768 | 0 | 0 | 0
  Serogroup C: >=1:65536: number analyzed (Participants) | 0 | 0 | 35
  Serogroup C: >=1:65536 |  |  | 0
  Serogroup Y: <1:4: number analyzed (Participants) | 32 | 26 | 35
  Serogroup Y: <1:4 | 3.1 | 11.5 | 94.3
  Serogroup Y: >=1:4: number analyzed (Participants) | 32 | 26 | 35
  Serogroup Y: >=1:4 | 96.9 | 88.5 | 5.7
  Serogroup Y: >=1:8: number analyzed (Participants) | 32 | 26 | 35
  Serogroup Y: >=1:8 | 93.8 | 73.1 | 5.7
  Serogroup Y: >=1:16: number analyzed (Participants) | 32 | 26 | 35
  Serogroup Y: >=1:16 | 78.1 | 34.6 | 2.9
  Serogroup Y: >=1:32: number analyzed (Participants) | 32 | 26 | 35
  Serogroup Y: >=1:32 | 50.0 | 19.2 | 2.9
  Serogroup Y: >=1:64: number analyzed (Participants) | 32 | 26 | 35
  Serogroup Y: >=1:64 | 28.1 | 11.5 | 2.9
  Serogroup Y: >=1:128: number analyzed (Participants) | 32 | 26 | 35
  Serogroup Y: >=1:128 | 12.5 | 3.8 | 2.9
  Serogroup Y: >=1:256: number analyzed (Participants) | 32 | 26 | 35
  Serogroup Y: >=1:256 | 6.3 | 0 | 2.9
  Serogroup Y: >=1:512: number analyzed (Participants) | 32 | 26 | 35
  Serogroup Y: >=1:512 | 0 | 0 | 0
  Serogroup Y: >=1:1024: number analyzed (Participants) | 32 | 26 | 35
  Serogroup Y: >=1:1024 | 0 | 0 | 0
  Serogroup Y: >=1:2048: number analyzed (Participants) | 32 | 26 | 35
  Serogroup Y: >=1:2048 | 0 | 0 | 0
  Serogroup Y: >=1:4096: number analyzed (Participants) | 32 | 26 | 35
  Serogroup Y: >=1:4096 | 0 | 0 | 0
  Serogroup Y: >=1:8192: number analyzed (Participants) | 32 | 26 | 35
  Serogroup Y: >=1:8192 | 0 | 0 | 0
  Serogroup Y: >=1:16384: number analyzed (Participants) | 32 | 26 | 35
  Serogroup Y: >=1:16384 | 0 | 0 | 0
  Serogroup Y: >=1:32768: number analyzed (Participants) | 32 | 26 | 35
  Serogroup Y: >=1:32768 | 0 | 0 | 0
  Serogroup Y: >=1:65536: number analyzed (Participants) | 0 | 0 | 35
  Serogroup Y: >=1:65536 |  |  | 0
  Serogroup W: <1:4 | 2.9 | 15.4 | 100
  Serogroup W: >=1:4 | 97.1 | 84.6 | 0
  Serogroup W: >=1:8 | 88.6 | 69.2 | 0
  Serogroup W: >=1:16 | 77.1 | 46.2 | 0
  Serogroup W: >=1:32 | 60.0 | 23.1 | 0
  Serogroup W: >=1:64 | 45.7 | 11.5 | 0
  Serogroup W: >=1:128 | 28.6 | 3.8 | 0
  Serogroup W: >=1:256 | 8.6 | 0 | 0
  Serogroup W: >=1:512 | 5.7 | 0 | 0
  Serogroup W: >=1:1024 | 0 | 0 | 0
  Serogroup W: >=1:2048 | 0 | 0 | 0
  Serogroup W: >=1:4096 | 0 | 0 | 0
  Serogroup W: >=1:8192 | 0 | 0 | 0
  Serogroup W: >=1:16384 | 0 | 0 | 0
  Serogroup W: >=1:32768 | 0 | 0 | 0
  Serogroup W: >=1:65536: number analyzed (Participants) | 0 | 0 | 35
  Serogroup W: >=1:65536 |  |  | 0

34. Secondary Outcome: Percentage of Participants With Distribution of hSBA Titers Against Meningococcal Serogroups A, C, Y, and W After Vaccination - PPAS3
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by hSBA assay. Percentage of participants with hSBA antibody titers distribution <1:4, >=1:4, >=1:8, >=1:16; >=1:32; >=1:64, >=1:128, >=1:256; >=1:512; >=1:1024; >=1:2048; >=1:4096; >=1:8192; >=1:16384; >=1:32768; >=1:65536 for meningococcal serogroups A, C, Y, and W were reported in this outcome measure.
Time Frame: 30 days post-vaccination at the age of 12 to 13 months (i.e., at the age of 13 to 14 months)
Population: Analysis was performed on PPAS3. Here, 'number analyzed' = participants with available data for each specified category and '0' in the number analyzed field denotes that no participant had available data for the specified titer category.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months) | Group 3: Bexsero® (2, 4, and 12 to 13 Months)
Number analyzed (Participants) | 178 | 169 | 86
percentage of participants
  Serogroup A: <1:4: number analyzed (Participants) | 159 | 156 | 80
  Serogroup A: <1:4 | 0 | 0 | 0
  Serogroup A: >=1:4: number analyzed (Participants) | 159 | 156 | 80
  Serogroup A: >=1:4 | 100 | 100 | 100
  Serogroup A: >=1:8: number analyzed (Participants) | 159 | 156 | 80
  Serogroup A: >=1:8 | 100 | 99.4 | 100
  Serogroup A: >=1:16: number analyzed (Participants) | 159 | 156 | 80
  Serogroup A: >=1:16 | 100 | 98.7 | 100
  Serogroup A: >=1:32: number analyzed (Participants) | 159 | 156 | 80
  Serogroup A: >=1:32 | 100 | 94.2 | 97.5
  Serogroup A: >=1:64: number analyzed (Participants) | 159 | 156 | 80
  Serogroup A: >=1:64 | 99.4 | 87.2 | 93.8
  Serogroup A: >=1:128: number analyzed (Participants) | 159 | 156 | 80
  Serogroup A: >=1:128 | 97.5 | 75.0 | 90.0
  Serogroup A: >=1:256: number analyzed (Participants) | 159 | 156 | 80
  Serogroup A: >=1:256 | 94.3 | 58.3 | 83.8
  Serogroup A: >=1:512: number analyzed (Participants) | 159 | 156 | 80
  Serogroup A: >=1:512 | 83.6 | 35.3 | 76.3
  Serogroup A: >=1:1024: number analyzed (Participants) | 159 | 156 | 80
  Serogroup A: >=1:1024 | 68.6 | 17.9 | 52.5
  Serogroup A: >=1:2048: number analyzed (Participants) | 159 | 156 | 80
  Serogroup A: >=1:2048 | 39.0 | 1.9 | 26.3
  Serogroup A: >=1:4096: number analyzed (Participants) | 159 | 156 | 80
  Serogroup A: >=1:4096 | 25.2 | 0 | 15.0
  Serogroup A: >=1:8192: number analyzed (Participants) | 159 | 156 | 80
  Serogroup A: >=1:8192 | 10.1 | 0 | 5.0
  Serogroup A: >=1:16384: number analyzed (Participants) | 159 | 156 | 80
  Serogroup A: >=1:16384 | 6.3 | 0 | 2.5
  Serogroup A: >=1:32768: number analyzed (Participants) | 159 | 156 | 80
  Serogroup A: >=1:32768 | 0.6 | 0 | 1.3
  Serogroup A: >=1:65536: number analyzed (Participants) | 0 | 0 | 80
  Serogroup A: >=1:65536 |  |  | 1.3
  Serogroup C: <1:4: number analyzed (Participants) | 168 | 165 | 85
  Serogroup C: <1:4 | 0 | 0 | 10.6
  Serogroup C: >=1:4: number analyzed (Participants) | 168 | 165 | 85
  Serogroup C: >=1:4 | 100 | 100 | 89.4
  Serogroup C: >=1:8: number analyzed (Participants) | 168 | 165 | 85
  Serogroup C: >=1:8 | 100 | 100 | 78.8
  Serogroup C: >=1:16: number analyzed (Participants) | 168 | 165 | 85
  Serogroup C: >=1:16 | 99.4 | 99.4 | 69.4
  Serogroup C: >=1:32: number analyzed (Participants) | 168 | 165 | 85
  Serogroup C: >=1:32 | 98.2 | 99.4 | 56.5
  Serogroup C: >=1:64: number analyzed (Participants) | 168 | 165 | 85
  Serogroup C: >=1:64 | 97.6 | 98.2 | 30.6
  Serogroup C: >=1:128: number analyzed (Participants) | 168 | 165 | 85
  Serogroup C: >=1:128 | 95.2 | 92.7 | 22.4
  Serogroup C: >=1:256: number analyzed (Participants) | 168 | 165 | 85
  Serogroup C: >=1:256 | 90.5 | 86.1 | 7.1
  Serogroup C: >=1:512: number analyzed (Participants) | 168 | 165 | 85
  Serogroup C: >=1:512 | 78.6 | 73.3 | 4.7
  Serogroup C: >=1:1024: number analyzed (Participants) | 168 | 165 | 85
  Serogroup C: >=1:1024 | 64.9 | 58.2 | 2.4
  Serogroup C: >=1:2048: number analyzed (Participants) | 168 | 165 | 85
  Serogroup C: >=1:2048 | 35.7 | 25.5 | 0
  Serogroup C: >=1:4096: number analyzed (Participants) | 168 | 165 | 85
  Serogroup C: >=1:4096 | 22.0 | 14.5 | 0
  Serogroup C: >=1:8192: number analyzed (Participants) | 168 | 165 | 85
  Serogroup C: >=1:8192 | 8.3 | 5.5 | 0
  Serogroup C: >=1:16384: number analyzed (Participants) | 168 | 165 | 85
  Serogroup C: >=1:16384 | 0.6 | 0.6 | 0
  Serogroup C: >=1:32768: number analyzed (Participants) | 168 | 165 | 85
  Serogroup C: >=1:32768 | 0 | 0.6 | 0
  Serogroup C: >=1:65536: number analyzed (Participants) | 0 | 0 | 85
  Serogroup C: >=1:65536 |  |  | 0
  Serogroup Y: <1:4: number analyzed (Participants) | 161 | 159 | 82
  Serogroup Y: <1:4 | 0 | 0 | 46.3
  Serogroup Y: >=1:4: number analyzed (Participants) | 161 | 159 | 82
  Serogroup Y: >=1:4 | 100 | 100 | 53.7
  Serogroup Y: >=1:8: number analyzed (Participants) | 161 | 159 | 82
  Serogroup Y: >=1:8 | 100 | 100 | 35.4
  Serogroup Y: >=1:16: number analyzed (Participants) | 161 | 159 | 82
  Serogroup Y: >=1:16 | 99.4 | 99.4 | 23.2
  Serogroup Y: >=1:32: number analyzed (Participants) | 161 | 159 | 82
  Serogroup Y: >=1:32 | 98.8 | 98.1 | 6.1
  Serogroup Y: >=1:64: number analyzed (Participants) | 161 | 159 | 82
  Serogroup Y: >=1:64 | 94.4 | 95.6 | 0
  Serogroup Y: >=1:128: number analyzed (Participants) | 161 | 159 | 82
  Serogroup Y: >=1:128 | 89.4 | 89.9 | 0
  Serogroup Y: >=1:256: number analyzed (Participants) | 161 | 159 | 82
  Serogroup Y: >=1:256 | 77.6 | 81.1 | 0
  Serogroup Y: >=1:512: number analyzed (Participants) | 161 | 159 | 82
  Serogroup Y: >=1:512 | 65.2 | 61.0 | 0
  Serogroup Y: >=1:1024: number analyzed (Participants) | 161 | 159 | 82
  Serogroup Y: >=1:1024 | 39.1 | 32.7 | 0
  Serogroup Y: >=1:2048: number analyzed (Participants) | 161 | 159 | 82
  Serogroup Y: >=1:2048 | 11.2 | 9.4 | 0
  Serogroup Y: >=1:4096: number analyzed (Participants) | 161 | 159 | 82
  Serogroup Y: >=1:4096 | 5.6 | 5.7 | 0
  Serogroup Y: >=1:8192: number analyzed (Participants) | 161 | 159 | 82
  Serogroup Y: >=1:8192 | 1.9 | 3.1 | 0
  Serogroup Y: >=1:16384: number analyzed (Participants) | 161 | 159 | 82
  Serogroup Y: >=1:16384 | 0 | 0 | 0
  Serogroup Y: >=1:32768: number analyzed (Participants) | 161 | 159 | 82
  Serogroup Y: >=1:32768 | 0 | 0 | 0
  Serogroup Y: >=1:65536: number analyzed (Participants) | 0 | 0 | 82
  Serogroup Y: >=1:65536 |  |  | 0
  Serogroup W: <1:4: number analyzed (Participants) | 172 | 160 | 86
  Serogroup W: <1:4 | 0.6 | 0 | 96.5
  Serogroup W: >=1:4: number analyzed (Participants) | 172 | 160 | 86
  Serogroup W: >=1:4 | 99.4 | 100 | 3.5
  Serogroup W: >=1:8: number analyzed (Participants) | 172 | 160 | 86
  Serogroup W: >=1:8 | 99.4 | 100 | 2.3
  Serogroup W: >=1:16: number analyzed (Participants) | 172 | 160 | 86
  Serogroup W: >=1:16 | 98.8 | 99.4 | 0
  Serogroup W: >=1:32: number analyzed (Participants) | 172 | 160 | 86
  Serogroup W: >=1:32 | 98.3 | 98.8 | 0
  Serogroup W: >=1:64: number analyzed (Participants) | 172 | 160 | 86
  Serogroup W: >=1:64 | 98.3 | 98.1 | 0
  Serogroup W: >=1:128: number analyzed (Participants) | 172 | 160 | 86
  Serogroup W: >=1:128 | 93.6 | 93.1 | 0
  Serogroup W: >=1:256: number analyzed (Participants) | 172 | 160 | 86
  Serogroup W: >=1:256 | 84.9 | 85.0 | 0
  Serogroup W: >=1:512: number analyzed (Participants) | 172 | 160 | 86
  Serogroup W: >=1:512 | 70.3 | 64.4 | 0
  Serogroup W: >=1:1024: number analyzed (Participants) | 172 | 160 | 86
  Serogroup W: >=1:1024 | 45.9 | 43.8 | 0
  Serogroup W: >=1:2048: number analyzed (Participants) | 172 | 160 | 86
  Serogroup W: >=1:2048 | 15.7 | 13.1 | 0
  Serogroup W: >=1:4096: number analyzed (Participants) | 172 | 160 | 86
  Serogroup W: >=1:4096 | 9.3 | 4.4 | 0
  Serogroup W: >=1:8192: number analyzed (Participants) | 172 | 160 | 86
  Serogroup W: >=1:8192 | 2.3 | 1.9 | 0
  Serogroup W: >=1:16384: number analyzed (Participants) | 172 | 160 | 86
  Serogroup W: >=1:16384 | 1.2 | 1.3 | 0
  Serogroup W: >=1:32768: number analyzed (Participants) | 172 | 160 | 86
  Serogroup W: >=1:32768 | 0 | 1.3 | 0
  Serogroup W: >=1:65536: number analyzed (Participants) | 0 | 0 | 86
  Serogroup W: >=1:65536 |  |  | 0

35. Secondary Outcome: Percentage of Participants With Distribution of rSBA Titers Against Meningococcal Serogroups A, C, Y, and W Before Vaccination - PPAS1
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by rSBA assay. Infancy was defined as up to 4 months of age. Percentage of participants with rSBA antibody titers distribution <1:4, >=1:4, >=1:8, >=1:16; >=1:32; >=1:64, >=1:128, >=1:256; >=1:512; >=1:1024; >=1:2048; >=1:4096; >=1:8192 for meningococcal serogroups A, C, Y, and W were reported in this outcome measure.
Time Frame: Before vaccination at the age of 3 months
Population: Analysis was performed on PPAS1. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified category. Here, '0' in the number analyzed field denotes that no participant had available data for the specified titer category.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months) | Group 3: Bexsero® (2, 4, and 12 to 13 Months)
Number analyzed (Participants) | 47 | 51 | 56
percentage of participants
  Serogroup A: <1:4: number analyzed (Participants) | 16 | 22 | 25
  Serogroup A: <1:4 | 100 | 100 | 100
  Serogroup A: >=1:4: number analyzed (Participants) | 16 | 22 | 25
  Serogroup A: >=1:4 | 0 | 0 | 0
  Serogroup A: >=1:8: number analyzed (Participants) | 16 | 22 | 25
  Serogroup A: >=1:8 | 0 | 0 | 0
  Serogroup A: >=1:16: number analyzed (Participants) | 16 | 22 | 25
  Serogroup A: >=1:16 | 0 | 0 | 0
  Serogroup A: >=1:32: number analyzed (Participants) | 16 | 22 | 25
  Serogroup A: >=1:32 | 0 | 0 | 0
  Serogroup A: >=1:64: number analyzed (Participants) | 16 | 22 | 25
  Serogroup A: >=1:64 | 0 | 0 | 0
  Serogroup A: >=1:128: number analyzed (Participants) | 16 | 22 | 25
  Serogroup A: >=1:128 | 0 | 0 | 0
  Serogroup A: >=1:256: number analyzed (Participants) | 16 | 22 | 25
  Serogroup A: >=1:256 | 0 | 0 | 0
  Serogroup A: >=1:512: number analyzed (Participants) | 16 | 22 | 25
  Serogroup A: >=1:512 | 0 | 0 | 0
  Serogroup A: >=1:1024: number analyzed (Participants) | 16 | 22 | 25
  Serogroup A: >=1:1024 | 0 | 0 | 0
  Serogroup A: >=1:2048: number analyzed (Participants) | 16 | 22 | 25
  Serogroup A: >=1:2048 | 0 | 0 | 0
  Serogroup A: >=1:4096: number analyzed (Participants) | 16 | 22 | 0
  Serogroup A: >=1:4096 | 0 | 0 |
  Serogroup A: >=1:8192: number analyzed (Participants) | 16 | 22 | 0
  Serogroup A: >=1:8192 | 0 | 0 |
  Serogroup C: <1:4: number analyzed (Participants) | 19 | 23 | 26
  Serogroup C: <1:4 | 84.2 | 82.6 | 84.6
  Serogroup C: >=1:4: number analyzed (Participants) | 19 | 23 | 26
  Serogroup C: >=1:4 | 15.8 | 17.4 | 15.4
  Serogroup C: >=1:8: number analyzed (Participants) | 19 | 23 | 26
  Serogroup C: >=1:8 | 15.8 | 17.4 | 11.5
  Serogroup C: >=1:16: number analyzed (Participants) | 19 | 23 | 26
  Serogroup C: >=1:16 | 10.5 | 17.4 | 7.7
  Serogroup C: >=1:32: number analyzed (Participants) | 19 | 23 | 26
  Serogroup C: >=1:32 | 5.3 | 17.4 | 0
  Serogroup C: >=1:64: number analyzed (Participants) | 19 | 23 | 26
  Serogroup C: >=1:64 | 5.3 | 13.0 | 0
  Serogroup C: >=1:128: number analyzed (Participants) | 19 | 23 | 26
  Serogroup C: >=1:128 | 0 | 4.3 | 0
  Serogroup C: >=1:256: number analyzed (Participants) | 19 | 23 | 26
  Serogroup C: >=1:256 | 0 | 4.3 | 0
  Serogroup C: >=1:512: number analyzed (Participants) | 19 | 23 | 26
  Serogroup C: >=1:512 | 0 | 0 | 0
  Serogroup C: >=1:1024: number analyzed (Participants) | 19 | 23 | 26
  Serogroup C: >=1:1024 | 0 | 0 | 0
  Serogroup C: >=1:2048: number analyzed (Participants) | 19 | 23 | 26
  Serogroup C: >=1:2048 | 0 | 0 | 0
  Serogroup C: >=1:4096: number analyzed (Participants) | 19 | 23 | 0
  Serogroup C: >=1:4096 | 0 | 0 |
  Serogroup C: >=1:8192: number analyzed (Participants) | 19 | 23 | 0
  Serogroup C: >=1:8192 | 0 | 0 |
  Serogroup Y: <1:4: number analyzed (Participants) | 19 | 23 | 26
  Serogroup Y: <1:4 | 89.5 | 87.0 | 84.6
  Serogroup Y: >=1:4: number analyzed (Participants) | 19 | 23 | 26
  Serogroup Y: >=1:4 | 10.5 | 13.0 | 15.4
  Serogroup Y: >=1:8: number analyzed (Participants) | 19 | 23 | 26
  Serogroup Y: >=1:8 | 10.5 | 13.0 | 15.4
  Serogroup Y: >=1:16: number analyzed (Participants) | 19 | 23 | 26
  Serogroup Y: >=1:16 | 10.5 | 8.7 | 7.7
  Serogroup Y: >=1:32: number analyzed (Participants) | 19 | 23 | 26
  Serogroup Y: >=1:32 | 10.5 | 4.3 | 3.8
  Serogroup Y: >=1:64: number analyzed (Participants) | 19 | 23 | 26
  Serogroup Y: >=1:64 | 0 | 4.3 | 3.8
  Serogroup Y: >=1:128: number analyzed (Participants) | 19 | 23 | 26
  Serogroup Y: >=1:128 | 0 | 0 | 0
  Serogroup Y: >=1:256: number analyzed (Participants) | 19 | 23 | 26
  Serogroup Y: >=1:256 | 0 | 0 | 0
  Serogroup Y: >=1:512: number analyzed (Participants) | 19 | 23 | 26
  Serogroup Y: >=1:512 | 0 | 0 | 0
  Serogroup Y: >=1:1024: number analyzed (Participants) | 19 | 23 | 26
  Serogroup Y: >=1:1024 | 0 | 0 | 0
  Serogroup Y: >=1:2048: number analyzed (Participants) | 19 | 23 | 26
  Serogroup Y: >=1:2048 | 0 | 0 | 0
  Serogroup Y: >=1:4096: number analyzed (Participants) | 19 | 23 | 0
  Serogroup Y: >=1:4096 | 0 | 0 |
  Serogroup Y: >=1:8192: number analyzed (Participants) | 19 | 23 | 0
  Serogroup Y: >=1:8192 | 0 | 0 |
  Serogroup W: <1:4: number analyzed (Participants) | 17 | 23 | 26
  Serogroup W: <1:4 | 88.2 | 100 | 96.2
  Serogroup W: >=1:4: number analyzed (Participants) | 17 | 23 | 26
  Serogroup W: >=1:4 | 11.8 | 0 | 3.8
  Serogroup W: >=1:8: number analyzed (Participants) | 17 | 23 | 26
  Serogroup W: >=1:8 | 11.8 | 0 | 3.8
  Serogroup W: >=1:16: number analyzed (Participants) | 17 | 23 | 26
  Serogroup W: >=1:16 | 11.8 | 0 | 3.8
  Serogroup W: >=1:32: number analyzed (Participants) | 17 | 23 | 26
  Serogroup W: >=1:32 | 11.8 | 0 | 3.8
  Serogroup W: >=1:64: number analyzed (Participants) | 17 | 23 | 26
  Serogroup W: >=1:64 | 5.9 | 0 | 3.8
  Serogroup W: >=1:128: number analyzed (Participants) | 17 | 23 | 26
  Serogroup W: >=1:128 | 0 | 0 | 0
  Serogroup W: >=1:256: number analyzed (Participants) | 17 | 23 | 26
  Serogroup W: >=1:256 | 0 | 0 | 0
  Serogroup W: >=1:512: number analyzed (Participants) | 17 | 23 | 26
  Serogroup W: >=1:512 | 0 | 0 | 0
  Serogroup W: >=1:1024: number analyzed (Participants) | 17 | 23 | 26
  Serogroup W: >=1:1024 | 0 | 0 | 0
  Serogroup W: >=1:2048: number analyzed (Participants) | 17 | 23 | 26
  Serogroup W: >=1:2048 | 0 | 0 | 0
  Serogroup W: >=1:4096: number analyzed (Participants) | 17 | 23 | 0
  Serogroup W: >=1:4096 | 0 | 0 |
  Serogroup W: >=1:8192: number analyzed (Participants) | 17 | 23 | 0
  Serogroup W: >=1:8192 | 0 | 0 |

36. Secondary Outcome: Percentage of Participants With Distribution of rSBA Titers Against Meningococcal Serogroups A, C, Y, and W After Vaccination - PPAS1
Description: as for outcome 35
Time Frame: 30 days post-vaccination at the age of 3 months (i.e., at the age of 4 months)
Population: as for outcome 35
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months) | Group 3: Bexsero® (2, 4, and 12 to 13 Months)
Number analyzed (Participants) | 47 | 51 | 56
percentage of participants
  Serogroup A: <1:4: number analyzed (Participants) | 36 | 32 | 36
  Serogroup A: <1:4 | 38.9 | 21.9 | 97.2
  Serogroup A: >=1:4: number analyzed (Participants) | 36 | 32 | 36
  Serogroup A: >=1:4 | 61.1 | 78.1 | 2.8
  Serogroup A: >=1:8: number analyzed (Participants) | 36 | 32 | 36
  Serogroup A: >=1:8 | 52.8 | 65.6 | 0
  Serogroup A: >=1:16: number analyzed (Participants) | 36 | 32 | 36
  Serogroup A: >=1:16 | 44.4 | 53.1 | 0
  Serogroup A: >=1:32: number analyzed (Participants) | 36 | 32 | 36
  Serogroup A: >=1:32 | 41.7 | 43.8 | 0
  Serogroup A: >=1:64: number analyzed (Participants) | 36 | 32 | 36
  Serogroup A: >=1:64 | 36.1 | 31.3 | 0
  Serogroup A: >=1:128: number analyzed (Participants) | 36 | 32 | 36
  Serogroup A: >=1:128 | 19.4 | 28.1 | 0
  Serogroup A: >=1:256: number analyzed (Participants) | 36 | 32 | 36
  Serogroup A: >=1:256 | 8.3 | 21.9 | 0
  Serogroup A: >=1:512: number analyzed (Participants) | 36 | 32 | 36
  Serogroup A: >=1:512 | 5.6 | 9.4 | 0
  Serogroup A: >=1:1024: number analyzed (Participants) | 36 | 32 | 36
  Serogroup A: >=1:1024 | 5.6 | 3.1 | 0
  Serogroup A: >=1:2048: number analyzed (Participants) | 36 | 32 | 36
  Serogroup A: >=1:2048 | 2.8 | 3.1 | 0
  Serogroup A: >=1:4096: number analyzed (Participants) | 36 | 32 | 0
  Serogroup A: >=1:4096 | 0 | 0 |
  Serogroup A: >=1:8192: number analyzed (Participants) | 36 | 32 | 0
  Serogroup A: >=1:8192 | 0 | 0 |
  Serogroup C: <1:4: number analyzed (Participants) | 38 | 32 | 37
  Serogroup C: <1:4 | 2.6 | 0 | 86.5
  Serogroup C: >=1:4: number analyzed (Participants) | 38 | 32 | 37
  Serogroup C: >=1:4 | 97.4 | 100 | 13.5
  Serogroup C: >=1:8: number analyzed (Participants) | 38 | 32 | 37
  Serogroup C: >=1:8 | 97.4 | 100 | 8.1
  Serogroup C: >=1:16: number analyzed (Participants) | 38 | 32 | 37
  Serogroup C: >=1:16 | 94.7 | 100 | 5.4
  Serogroup C: >=1:32: number analyzed (Participants) | 38 | 32 | 37
  Serogroup C: >=1:32 | 89.5 | 100 | 5.4
  Serogroup C: >=1:64: number analyzed (Participants) | 38 | 32 | 37
  Serogroup C: >=1:64 | 81.6 | 96.9 | 0
  Serogroup C: >=1:128: number analyzed (Participants) | 38 | 32 | 37
  Serogroup C: >=1:128 | 78.9 | 96.9 | 0
  Serogroup C: >=1:256: number analyzed (Participants) | 38 | 32 | 37
  Serogroup C: >=1:256 | 71.1 | 65.6 | 0
  Serogroup C: >=1:512: number analyzed (Participants) | 38 | 32 | 37
  Serogroup C: >=1:512 | 55.3 | 40.6 | 0
  Serogroup C: >=1:1024: number analyzed (Participants) | 38 | 32 | 37
  Serogroup C: >=1:1024 | 23.7 | 28.1 | 0
  Serogroup C: >=1:2048: number analyzed (Participants) | 38 | 32 | 37
  Serogroup C: >=1:2048 | 5.3 | 9.4 | 0
  Serogroup C: >=1:4096: number analyzed (Participants) | 38 | 32 | 0
  Serogroup C: >=1:4096 | 2.6 | 3.1 |
  Serogroup C: >=1:8192: number analyzed (Participants) | 38 | 32 | 0
  Serogroup C: >=1:8192 | 0 | 3.1 |
  Serogroup Y: <1:4: number analyzed (Participants) | 36 | 25 | 31
  Serogroup Y: <1:4 | 8.3 | 8.0 | 90.3
  Serogroup Y: >=1:4: number analyzed (Participants) | 36 | 25 | 31
  Serogroup Y: >=1:4 | 91.7 | 92.0 | 9.7
  Serogroup Y: >=1:8: number analyzed (Participants) | 36 | 25 | 31
  Serogroup Y: >=1:8 | 91.7 | 92.0 | 9.7
  Serogroup Y: >=1:16: number analyzed (Participants) | 36 | 25 | 31
  Serogroup Y: >=1:16 | 88.9 | 88.0 | 9.7
  Serogroup Y: >=1:32: number analyzed (Participants) | 36 | 25 | 31
  Serogroup Y: >=1:32 | 83.3 | 80.0 | 6.5
  Serogroup Y: >=1:64: number analyzed (Participants) | 36 | 25 | 31
  Serogroup Y: >=1:64 | 80.6 | 72.0 | 3.2
  Serogroup Y: >=1:128: number analyzed (Participants) | 36 | 25 | 31
  Serogroup Y: >=1:128 | 80.6 | 68.0 | 3.2
  Serogroup Y: >=1:256: number analyzed (Participants) | 36 | 25 | 31
  Serogroup Y: >=1:256 | 63.9 | 48.0 | 3.2
  Serogroup Y: >=1:512: number analyzed (Participants) | 36 | 25 | 31
  Serogroup Y: >=1:512 | 36.1 | 36.0 | 3.2
  Serogroup Y: >=1:1024: number analyzed (Participants) | 36 | 25 | 31
  Serogroup Y: >=1:1024 | 5.6 | 12.0 | 3.2
  Serogroup Y: >=1:2048: number analyzed (Participants) | 36 | 25 | 31
  Serogroup Y: >=1:2048 | 2.8 | 4.0 | 3.2
  Serogroup Y: >=1:4096: number analyzed (Participants) | 36 | 25 | 0
  Serogroup Y: >=1:4096 | 0 | 4.0 |
  Serogroup Y: >=1:8192: number analyzed (Participants) | 36 | 25 | 0
  Serogroup Y: >=1:8192 | 0 | 0 |
  Serogroup W: <1:4: number analyzed (Participants) | 36 | 30 | 36
  Serogroup W: <1:4 | 22.2 | 33.3 | 100
  Serogroup W: >=1:4: number analyzed (Participants) | 36 | 30 | 36
  Serogroup W: >=1:4 | 77.8 | 66.7 | 0
  Serogroup W: >=1:8: number analyzed (Participants) | 36 | 30 | 36
  Serogroup W: >=1:8 | 77.8 | 63.3 | 0
  Serogroup W: >=1:16: number analyzed (Participants) | 36 | 30 | 36
  Serogroup W: >=1:16 | 77.8 | 63.3 | 0
  Serogroup W: >=1:32: number analyzed (Participants) | 36 | 30 | 36
  Serogroup W: >=1:32 | 75.0 | 63.3 | 0
  Serogroup W: >=1:64: number analyzed (Participants) | 36 | 30 | 36
  Serogroup W: >=1:64 | 75.0 | 63.3 | 0
  Serogroup W: >=1:128: number analyzed (Participants) | 36 | 30 | 36
  Serogroup W: >=1:128 | 75.0 | 53.3 | 0
  Serogroup W: >=1:256: number analyzed (Participants) | 36 | 30 | 36
  Serogroup W: >=1:256 | 50.0 | 50.0 | 0
  Serogroup W: >=1:512: number analyzed (Participants) | 36 | 30 | 36
  Serogroup W: >=1:512 | 19.4 | 26.7 | 0
  Serogroup W: >=1:1024: number analyzed (Participants) | 36 | 30 | 36
  Serogroup W: >=1:1024 | 11.1 | 13.3 | 0
  Serogroup W: >=1:2048: number analyzed (Participants) | 36 | 30 | 36
  Serogroup W: >=1:2048 | 5.6 | 3.3 | 0
  Serogroup W: >=1:4096: number analyzed (Participants) | 36 | 30 | 0
  Serogroup W: >=1:4096 | 0 | 0 |
  Serogroup W: >=1:8192: number analyzed (Participants) | 36 | 30 | 0
  Serogroup W: >=1:8192 | 0 | 0 |

37. Secondary Outcome: Percentage of Participants With Distribution of rSBA Titers Against Meningococcal Serogroups A, C, Y, and W Before Vaccination - PPAS3
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by rSBA assay. Infancy was defined as up to 4 months of age. Percentage of participants with rSBA antibody titers distribution <1:4, >=1:4, >=1:8, >=1:16; >=1:32; >=1:64, >=1:128, >=1:256; >=1:512; >=1:1024; >=1:2048; >=1:4096; >=1:8192; >=1:16384; >=1:32768 for meningococcal serogroups A, C, Y, and W were reported in this outcome measure.
Time Frame: Before vaccination at the age of 12 to 13 months
Population: as for outcome 33
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months) | Group 3: Bexsero® (2, 4, and 12 to 13 Months)
Number analyzed (Participants) | 7 | 5 | 6
percentage of participants
  Serogroup A: <1:4: number analyzed (Participants) | 6 | 5 | 6
  Serogroup A: <1:4 | 50.0 | 20.0 | 50.0
  Serogroup A: >=1:4: number analyzed (Participants) | 6 | 5 | 6
  Serogroup A: >=1:4 | 50.0 | 80.0 | 50.0
  Serogroup A: >=1:8: number analyzed (Participants) | 6 | 5 | 6
  Serogroup A: >=1:8 | 50.0 | 80.0 | 50.0
  Serogroup A: >=1:16: number analyzed (Participants) | 6 | 5 | 6
  Serogroup A: >=1:16 | 50.0 | 80.0 | 50.0
  Serogroup A: >=1:32: number analyzed (Participants) | 6 | 5 | 6
  Serogroup A: >=1:32 | 50.0 | 80.0 | 50.0
  Serogroup A: >=1:64: number analyzed (Participants) | 6 | 5 | 6
  Serogroup A: >=1:64 | 50.0 | 80.0 | 50.0
  Serogroup A: >=1:128: number analyzed (Participants) | 6 | 5 | 6
  Serogroup A: >=1:128 | 50.0 | 80.0 | 33.3
  Serogroup A: >=1:256: number analyzed (Participants) | 6 | 5 | 6
  Serogroup A: >=1:256 | 33.3 | 60.0 | 33.3
  Serogroup A: >=1:512: number analyzed (Participants) | 6 | 5 | 6
  Serogroup A: >=1:512 | 33.3 | 40.0 | 33.3
  Serogroup A: >=1:1024: number analyzed (Participants) | 6 | 5 | 6
  Serogroup A: >=1:1024 | 33.3 | 40.0 | 16.7
  Serogroup A: >=1:2048: number analyzed (Participants) | 6 | 5 | 6
  Serogroup A: >=1:2048 | 0 | 20.0 | 16.7
  Serogroup A: >=1:4096: number analyzed (Participants) | 6 | 5 | 6
  Serogroup A: >=1:4096 | 0 | 0 | 16.7
  Serogroup A: >=1:8192: number analyzed (Participants) | 6 | 5 | 0
  Serogroup A: >=1:8192 | 0 | 0 |
  Serogroup A: >=1:16384: number analyzed (Participants) | 6 | 5 | 0
  Serogroup A: >=1:16384 | 0 | 0 |
  Serogroup A: >=1:32768: number analyzed (Participants) | 6 | 5 | 0
  Serogroup A: >=1:32768 | 0 | 0 |
  Serogroup C: <1:4 | 0 | 80.0 | 100
  Serogroup C: >=1:4 | 100 | 20.0 | 0
  Serogroup C: >=1:8 | 100 | 20.0 | 0
  Serogroup C: >=1:16 | 85.7 | 20.0 | 0
  Serogroup C: >=1:32 | 71.4 | 20.0 | 0
  Serogroup C: >=1:64 | 71.4 | 0 | 0
  Serogroup C: >=1:128 | 42.9 | 0 | 0
  Serogroup C: >=1:256 | 14.3 | 0 | 0
  Serogroup C: >=1:512 | 0 | 0 | 0
  Serogroup C: >=1:1024 | 0 | 0 | 0
  Serogroup C: >=1:2048 | 0 | 0 | 0
  Serogroup C: >=1:4096 | 0 | 0 | 0
  Serogroup C: >=1:8192: number analyzed (Participants) | 7 | 5 | 0
  Serogroup C: >=1:8192 | 0 | 0 |
  Serogroup C: >=1:16384: number analyzed (Participants) | 7 | 5 | 0
  Serogroup C: >=1:16384 | 0 | 0 |
  Serogroup C: >=1:32768: number analyzed (Participants) | 7 | 5 | 0
  Serogroup C: >=1:32768 | 0 | 0 |
  Serogroup Y: <1:4 | 14.3 | 40.0 | 100
  Serogroup Y: >=1:4 | 85.7 | 60.0 | 0
  Serogroup Y: >=1:8 | 85.7 | 40.0 | 0
  Serogroup Y: >=1:16 | 85.7 | 40.0 | 0
  Serogroup Y: >=1:32 | 71.4 | 20.0 | 0
  Serogroup Y: >=1:64 | 57.1 | 20.0 | 0
  Serogroup Y: >=1:128 | 28.6 | 0 | 0
  Serogroup Y: >=1:256 | 14.3 | 0 | 0
  Serogroup Y: >=1:512 | 14.3 | 0 | 0
  Serogroup Y: >=1:1024 | 14.3 | 0 | 0
  Serogroup Y: >=1:2048 | 14.3 | 0 | 0
  Serogroup Y: >=1:4096 | 14.3 | 0 | 0
  Serogroup Y: >=1:8192: number analyzed (Participants) | 7 | 5 | 0
  Serogroup Y: >=1:8192 | 0 | 0 |
  Serogroup Y: >=1:16384: number analyzed (Participants) | 7 | 5 | 0
  Serogroup Y: >=1:16384 | 0 | 0 |
  Serogroup Y: >=1:32768: number analyzed (Participants) | 7 | 5 | 0
  Serogroup Y: >=1:32768 | 0 | 0 |
  Serogroup W: <1:4: number analyzed (Participants) | 5 | 5 | 6
  Serogroup W: <1:4 | 40.0 | 40.0 | 100
  Serogroup W: >=1:4: number analyzed (Participants) | 5 | 5 | 6
  Serogroup W: >=1:4 | 60.0 | 60.0 | 0
  Serogroup W: >=1:8: number analyzed (Participants) | 5 | 5 | 6
  Serogroup W: >=1:8 | 40.0 | 60.0 | 0
  Serogroup W: >=1:16: number analyzed (Participants) | 5 | 5 | 6
  Serogroup W: >=1:16 | 40.0 | 40.0 | 0
  Serogroup W: >=1:32: number analyzed (Participants) | 5 | 5 | 6
  Serogroup W: >=1:32 | 20.0 | 20.0 | 0
  Serogroup W: >=1:64: number analyzed (Participants) | 5 | 5 | 6
  Serogroup W: >=1:64 | 20.0 | 20.0 | 0
  Serogroup W: >=1:128: number analyzed (Participants) | 5 | 5 | 6
  Serogroup W: >=1:128 | 20.0 | 0 | 0
  Serogroup W: >=1:256: number analyzed (Participants) | 5 | 5 | 6
  Serogroup W: >=1:256 | 0 | 0 | 0
  Serogroup W: >=1:512: number analyzed (Participants) | 5 | 5 | 6
  Serogroup W: >=1:512 | 0 | 0 | 0
  Serogroup W: >=1:1024: number analyzed (Participants) | 5 | 5 | 6
  Serogroup W: >=1:1024 | 0 | 0 | 0
  Serogroup W: >=1:2048: number analyzed (Participants) | 5 | 5 | 6
  Serogroup W: >=1:2048 | 0 | 0 | 0
  Serogroup W: >=1:4096: number analyzed (Participants) | 5 | 5 | 6
  Serogroup W: >=1:4096 | 0 | 0 | 0
  Serogroup W: >=1:8192: number analyzed (Participants) | 5 | 5 | 0
  Serogroup W: >=1:8192 | 0 | 0 |
  Serogroup W: >=1:16384: number analyzed (Participants) | 5 | 5 | 0
  Serogroup W: >=1:16384 | 0 | 0 |
  Serogroup W: >=1:32768: number analyzed (Participants) | 5 | 5 | 0
  Serogroup W: >=1:32768 | 0 | 0 |

38. Secondary Outcome: Percentage of Participants With Distribution of rSBA Titers Against Meningococcal Serogroups A, C, Y, and W After Vaccination - PPAS3
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by rSBA assay. Percentage of participants with rSBA antibody titers distribution <1:4, >=1:4, >=1:8, >=1:16; >=1:32; >=1:64, >=1:128, >=1:256; >=1:512; >=1:1024; >=1:2048; >=1:4096; >=1:8192; >=1:16384; >=1:32768 for meningococcal serogroups A, C, Y, and W were reported in this outcome measure.
Time Frame: 30 days post-vaccination at the age of 12 to 13 months (i.e., at the age of 13 to 14 months)
Population: as for outcome 33
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months) | Group 3: Bexsero® (2, 4, and 12 to 13 Months)
Number analyzed (Participants) | 54 | 54 | 52
percentage of participants
  Serogroup A: <1:4: number analyzed (Participants) | 47 | 43 | 41
  Serogroup A: <1:4 | 0 | 0 | 14.6
  Serogroup A: >=1:4: number analyzed (Participants) | 47 | 43 | 41
  Serogroup A: >=1:4 | 100 | 100 | 85.4
  Serogroup A: >=1:8: number analyzed (Participants) | 47 | 43 | 41
  Serogroup A: >=1:8 | 100 | 100 | 85.4
  Serogroup A: >=1:16: number analyzed (Participants) | 47 | 43 | 41
  Serogroup A: >=1:16 | 100 | 100 | 85.4
  Serogroup A: >=1:32: number analyzed (Participants) | 47 | 43 | 41
  Serogroup A: >=1:32 | 100 | 100 | 85.4
  Serogroup A: >=1:64: number analyzed (Participants) | 47 | 43 | 41
  Serogroup A: >=1:64 | 100 | 100 | 85.4
  Serogroup A: >=1:128: number analyzed (Participants) | 47 | 43 | 41
  Serogroup A: >=1:128 | 100 | 97.7 | 85.4
  Serogroup A: >=1:256: number analyzed (Participants) | 47 | 43 | 41
  Serogroup A: >=1:256 | 100 | 97.7 | 75.6
  Serogroup A: >=1:512: number analyzed (Participants) | 47 | 43 | 41
  Serogroup A: >=1:512 | 97.9 | 88.4 | 68.3
  Serogroup A: >=1:1024: number analyzed (Participants) | 47 | 43 | 41
  Serogroup A: >=1:1024 | 87.2 | 79.1 | 51.2
  Serogroup A: >=1:2048: number analyzed (Participants) | 47 | 43 | 41
  Serogroup A: >=1:2048 | 53.2 | 51.2 | 36.6
  Serogroup A: >=1:4096: number analyzed (Participants) | 47 | 43 | 41
  Serogroup A: >=1:4096 | 29.8 | 32.6 | 17.1
  Serogroup A: >=1:8192: number analyzed (Participants) | 47 | 43 | 0
  Serogroup A: >=1:8192 | 6.4 | 9.3 |
  Serogroup A: >=1:16384: number analyzed (Participants) | 47 | 43 | 0
  Serogroup A: >=1:16384 | 2.1 | 0 |
  Serogroup A: >=1:32768: number analyzed (Participants) | 47 | 43 | 0
  Serogroup A: >=1:32768 | 0 | 0 |
  Serogroup C: <1:4: number analyzed (Participants) | 47 | 43 | 44
  Serogroup C: <1:4 | 0 | 0 | 88.6
  Serogroup C: >=1:4: number analyzed (Participants) | 47 | 43 | 44
  Serogroup C: >=1:4 | 100 | 100 | 11.4
  Serogroup C: >=1:8: number analyzed (Participants) | 47 | 43 | 44
  Serogroup C: >=1:8 | 100 | 100 | 11.4
  Serogroup C: >=1:16: number analyzed (Participants) | 47 | 43 | 44
  Serogroup C: >=1:16 | 100 | 100 | 11.4
  Serogroup C: >=1:32: number analyzed (Participants) | 47 | 43 | 44
  Serogroup C: >=1:32 | 100 | 100 | 11.4
  Serogroup C: >=1:64: number analyzed (Participants) | 47 | 43 | 44
  Serogroup C: >=1:64 | 100 | 100 | 11.4
  Serogroup C: >=1:128: number analyzed (Participants) | 47 | 43 | 44
  Serogroup C: >=1:128 | 100 | 100 | 9.1
  Serogroup C: >=1:256: number analyzed (Participants) | 47 | 43 | 44
  Serogroup C: >=1:256 | 100 | 95.3 | 0
  Serogroup C: >=1:512: number analyzed (Participants) | 47 | 43 | 44
  Serogroup C: >=1:512 | 89.4 | 88.4 | 0
  Serogroup C: >=1:1024: number analyzed (Participants) | 47 | 43 | 44
  Serogroup C: >=1:1024 | 74.5 | 72.1 | 0
  Serogroup C: >=1:2048: number analyzed (Participants) | 47 | 43 | 44
  Serogroup C: >=1:2048 | 51.1 | 53.5 | 0
  Serogroup C: >=1:4096: number analyzed (Participants) | 47 | 43 | 44
  Serogroup C: >=1:4096 | 21.3 | 34.9 | 0
  Serogroup C: >=1:8192: number analyzed (Participants) | 47 | 43 | 0
  Serogroup C: >=1:8192 | 8.5 | 9.3 |
  Serogroup C: >=1:16384: number analyzed (Participants) | 47 | 43 | 0
  Serogroup C: >=1:16384 | 0 | 4.7 |
  Serogroup C: >=1:32768: number analyzed (Participants) | 47 | 43 | 0
  Serogroup C: >=1:32768 | 0 | 0 |
  Serogroup Y: <1:4: number analyzed (Participants) | 45 | 43 | 43
  Serogroup Y: <1:4 | 0 | 0 | 7.0
  Serogroup Y: >=1:4: number analyzed (Participants) | 45 | 43 | 43
  Serogroup Y: >=1:4 | 100 | 100 | 93.0
  Serogroup Y: >=1:8: number analyzed (Participants) | 45 | 43 | 43
  Serogroup Y: >=1:8 | 100 | 100 | 93.0
  Serogroup Y: >=1:16: number analyzed (Participants) | 45 | 43 | 43
  Serogroup Y: >=1:16 | 100 | 100 | 93.0
  Serogroup Y: >=1:32: number analyzed (Participants) | 45 | 43 | 43
  Serogroup Y: >=1:32 | 100 | 97.7 | 93.0
  Serogroup Y: >=1:64: number analyzed (Participants) | 45 | 43 | 43
  Serogroup Y: >=1:64 | 100 | 97.7 | 93.0
  Serogroup Y: >=1:128: number analyzed (Participants) | 45 | 43 | 43
  Serogroup Y: >=1:128 | 100 | 97.7 | 93.0
  Serogroup Y: >=1:256: number analyzed (Participants) | 45 | 43 | 43
  Serogroup Y: >=1:256 | 100 | 95.3 | 90.7
  Serogroup Y: >=1:512: number analyzed (Participants) | 45 | 43 | 43
  Serogroup Y: >=1:512 | 97.8 | 95.3 | 79.1
  Serogroup Y: >=1:1024: number analyzed (Participants) | 45 | 43 | 43
  Serogroup Y: >=1:1024 | 93.3 | 79.1 | 67.4
  Serogroup Y: >=1:2048: number analyzed (Participants) | 45 | 43 | 43
  Serogroup Y: >=1:2048 | 77.8 | 53.5 | 46.5
  Serogroup Y: >=1:4096: number analyzed (Participants) | 45 | 43 | 43
  Serogroup Y: >=1:4096 | 44.4 | 20.9 | 11.6
  Serogroup Y: >=1:8192: number analyzed (Participants) | 45 | 43 | 0
  Serogroup Y: >=1:8192 | 17.8 | 9.3 |
  Serogroup Y: >=1:16384: number analyzed (Participants) | 45 | 43 | 0
  Serogroup Y: >=1:16384 | 2.2 | 0 |
  Serogroup Y: >=1:32768: number analyzed (Participants) | 45 | 43 | 0
  Serogroup Y: >=1:32768 | 2.2 | 0 |
  Serogroup W: <1:4: number analyzed (Participants) | 46 | 43 | 42
  Serogroup W: <1:4 | 0 | 0 | 81.0
  Serogroup W: >=1:4: number analyzed (Participants) | 46 | 43 | 42
  Serogroup W: >=1:4 | 100 | 100 | 19.0
  Serogroup W: >=1:8: number analyzed (Participants) | 46 | 43 | 42
  Serogroup W: >=1:8 | 100 | 100 | 16.7
  Serogroup W: >=1:16: number analyzed (Participants) | 46 | 43 | 42
  Serogroup W: >=1:16 | 100 | 100 | 16.7
  Serogroup W: >=1:32: number analyzed (Participants) | 46 | 43 | 42
  Serogroup W: >=1:32 | 100 | 100 | 16.7
  Serogroup W: >=1:64: number analyzed (Participants) | 46 | 43 | 42
  Serogroup W: >=1:64 | 100 | 100 | 16.7
  Serogroup W: >=1:128: number analyzed (Participants) | 46 | 43 | 42
  Serogroup W: >=1:128 | 100 | 97.7 | 11.9
  Serogroup W: >=1:256: number analyzed (Participants) | 46 | 43 | 42
  Serogroup W: >=1:256 | 100 | 97.7 | 4.8
  Serogroup W: >=1:512: number analyzed (Participants) | 46 | 43 | 42
  Serogroup W: >=1:512 | 97.8 | 95.3 | 2.4
  Serogroup W: >=1:1024: number analyzed (Participants) | 46 | 43 | 42
  Serogroup W: >=1:1024 | 87.0 | 86.0 | 0
  Serogroup W: >=1:2048: number analyzed (Participants) | 46 | 43 | 42
  Serogroup W: >=1:2048 | 73.9 | 74.4 | 0
  Serogroup W: >=1:4096: number analyzed (Participants) | 46 | 43 | 42
  Serogroup W: >=1:4096 | 39.1 | 46.5 | 0
  Serogroup W: >=1:8192: number analyzed (Participants) | 46 | 43 | 0
  Serogroup W: >=1:8192 | 28.3 | 25.6 |
  Serogroup W: >=1:16384: number analyzed (Participants) | 46 | 43 | 0
  Serogroup W: >=1:16384 | 2.2 | 9.3 |
  Serogroup W: >=1:32768: number analyzed (Participants) | 46 | 43 | 0
  Serogroup W: >=1:32768 | 0 | 0 |

39. Secondary Outcome: Geometric Mean Titers of Antibodies Measured by hSBA Against Meningococcal Serogroups A, C, Y, and W: Group 1 and 2 - PPAS2
Description: as for outcome 2
Time Frame: 30 days post-vaccination at the age of 3 months (i.e., at the age of 4 months) and before vaccination at the age of 12-13 months
Population: Analysis was performed on per-protocol analysis set 2 (PPAS2) defined for accessing ACYW immune response data for participants who received at least 1 dose of study vaccine in infancy and had valid post-vaccination serology results at 12 to13 months of age, with no relevant protocol violations. Here, 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for Group 3.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 41 | 36
titers
  Serogroup A: 30 days after 3-month vaccination: number analyzed (Participants) | 27 | 28
  Serogroup A: 30 days after 3-month vaccination | 12.7 [8.68 to 18.6] | 9.28 [6.29 to 13.7]
  Serogroup A: Before 12-13 months vaccination: number analyzed (Participants) | 36 | 36
  Serogroup A: Before 12-13 months vaccination | 46.1 [28.9 to 73.6] | 31.4 [18.9 to 52.1]
  Serogroup C: 30 days after 3-month vaccination: number analyzed (Participants) | 28 | 28
  Serogroup C: 30 days after 3-month vaccination | 95.1 [54.1 to 167] | 59.4 [31.6 to 112]
  Serogroup C: Before 12-13 months vaccination | 24.4 [15.5 to 38.5] | 16.6 [9.71 to 28.5]
  Serogroup Y: 30 days after 3-month vaccination: number analyzed (Participants) | 29 | 26
  Serogroup Y: 30 days after 3-month vaccination | 9.69 [5.69 to 16.5] | 4.95 [3.39 to 7.22]
  Serogroup Y: Before 12-13 months vaccination: number analyzed (Participants) | 38 | 33
  Serogroup Y: Before 12-13 months vaccination | 21.4 [14.6 to 31.5] | 12.4 [8.36 to 18.5]
  Serogroup W: 30 days after 3-month vaccination: number analyzed (Participants) | 27 | 28
  Serogroup W: 30 days after 3-month vaccination | 4.32 [2.99 to 6.24] | 3.62 [2.60 to 5.05]
  Serogroup W: Before 12-13 months vaccination: number analyzed (Participants) | 41 | 35
  Serogroup W: Before 12-13 months vaccination | 29.4 [18.7 to 46.3] | 11.2 [7.59 to 16.5]

40. Secondary Outcome: Percentage of Participants With hSBA Antibody Titers >=1:4 and >=1:8 Against Meningococcal Serogroups A, C, Y, and W - PPAS2
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by hSBA assay. Percentage of participants with hSBA antibody titers >=1.4 and >=1:8 for meningococcal serogroups A, C, Y, and W were reported in this outcome measure.
Time Frame: as for outcome 39
Population: Analysis was performed on PPAS2. Here, 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for Group 3.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 41 | 36
percentage of participants
  Serogroup A: 30 days after 3-month vaccination: >= 1:4: number analyzed (Participants) | 27 | 28
  Serogroup A: 30 days after 3-month vaccination: >= 1:4 | 88.9 [70.8 to 97.6] | 89.3 [71.8 to 97.7]
  Serogroup A: 30 days after 3-month vaccination: >= 1:8: number analyzed (Participants) | 27 | 28
  Serogroup A: 30 days after 3-month vaccination: >= 1:8 | 81.5 [61.9 to 93.7] | 64.3 [44.1 to 81.4]
  Serogroup A: Before 12-13 months vaccination: >= 1:4: number analyzed (Participants) | 36 | 36
  Serogroup A: Before 12-13 months vaccination: >= 1:4 | 97.2 [85.5 to 99.9] | 97.2 [85.5 to 99.9]
  Serogroup A: Before 12-13 months vaccination: >= 1:8: number analyzed (Participants) | 36 | 36
  Serogroup A: Before 12-13 months vaccination: >= 1:8 | 91.7 [77.5 to 98.2] | 83.3 [67.2 to 93.6]
  Serogroup C: 30 days after 3-month vaccination: >= 1:4: number analyzed (Participants) | 28 | 28
  Serogroup C: 30 days after 3-month vaccination: >= 1:4 | 100 [87.7 to 100] | 96.4 [81.7 to 99.9]
  Serogroup C: 30 days after 3-month vaccination: >= 1:8: number analyzed (Participants) | 28 | 28
  Serogroup C: 30 days after 3-month vaccination: >= 1:8 | 92.9 [76.5 to 99.1] | 92.9 [76.5 to 99.1]
  Serogroup C: Before 12-13 months vaccination: >= 1:4 | 87.8 [73.8 to 95.9] | 80.6 [64.0 to 91.8]
  Serogroup C: Before 12-13 months vaccination: >= 1:8 | 80.5 [65.1 to 91.2] | 69.4 [51.9 to 83.7]
  Serogroup Y: 30 days after 3-month vaccination: >= 1:4: number analyzed (Participants) | 29 | 26
  Serogroup Y: 30 days after 3-month vaccination: >= 1:4 | 75.9 [56.5 to 89.7] | 57.7 [36.9 to 76.6]
  Serogroup Y: 30 days after 3-month vaccination: >= 1:8: number analyzed (Participants) | 29 | 26
  Serogroup Y: 30 days after 3-month vaccination: >= 1:8 | 65.5 [45.7 to 82.1] | 46.2 [26.6 to 66.6]
  Serogroup Y: Before 12-13 months vaccination: >= 1:4: number analyzed (Participants) | 38 | 33
  Serogroup Y: Before 12-13 months vaccination: >= 1:4 | 94.7 [82.3 to 99.4] | 90.9 [75.7 to 98.1]
  Serogroup Y: Before 12-13 months vaccination: >= 1:8: number analyzed (Participants) | 38 | 33
  Serogroup Y: Before 12-13 months vaccination: >= 1:8 | 89.5 [75.2 to 97.1] | 78.8 [61.1 to 91.0]
  Serogroup W: 30 days after 3-month vaccination: >= 1:4: number analyzed (Participants) | 27 | 28
  Serogroup W: 30 days after 3-month vaccination: >= 1:4 | 51.9 [31.9 to 71.3] | 39.3 [21.5 to 59.4]
  Serogroup W: 30 days after 3-month vaccination: >= 1:8: number analyzed (Participants) | 27 | 28
  Serogroup W: 30 days after 3-month vaccination: >= 1:8 | 37.0 [19.4 to 57.6] | 28.6 [13.2 to 48.7]
  Serogroup W: Before 12-13 months vaccination: >= 1:4: number analyzed (Participants) | 41 | 35
  Serogroup W: Before 12-13 months vaccination: >= 1:4 | 92.7 [80.1 to 98.5] | 88.6 [73.3 to 96.8]
  Serogroup W: Before 12-13 months vaccination: >= 1:8: number analyzed (Participants) | 41 | 35
  Serogroup W: Before 12-13 months vaccination: >= 1:8 | 85.4 [70.8 to 94.4] | 68.6 [50.7 to 83.1]

41. Secondary Outcome: Geometric Mean Titers of Antibodies Measured by rSBA Against Meningococcal Serogroups A, C, Y, and W: Group 1 and 2 - PPAS2
Description: as for outcome 9
Time Frame: as for outcome 39
Population: Analysis was performed on PPAS2. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for Group 3.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 11 | 10
titers
  Serogroup A: 30 days after 3-month vaccination: number analyzed (Participants) | 3 | 6
  Serogroup A: 30 days after 3-month vaccination | 80.6 [NA to NA] — 95% CI was not computable as the sample size was too small to compute valid data. | 18.0 [3.33 to 96.9]
  Serogroup A: Before 12-13 months vaccination: number analyzed (Participants) | 7 | 9
  Serogroup A: Before 12-13 months vaccination | 21.5 [1.29 to 360] | 27.4 [2.92 to 258]
  Serogroup C: 30 days after 3-month vaccination: number analyzed (Participants) | 4 | 6
  Serogroup C: 30 days after 3-month vaccination | 431 [NA to NA] — 95% CI was not computable as the sample size was too small to compute valid data. | 144 [44.8 to 461]
  Serogroup C: Before 12-13 months vaccination: number analyzed (Participants) | 8 | 9
  Serogroup C: Before 12-13 months vaccination | 38.1 [9.61 to 151] | 11.8 [1.96 to 70.4]
  Serogroup Y: 30 days after 3-month vaccination: number analyzed (Participants) | 3 | 6
  Serogroup Y: 30 days after 3-month vaccination | 323 [NA to NA] — 95% CI was not computable as the sample size was too small to compute valid data. | 102 [22.6 to 456]
  Serogroup Y: Before 12-13 months vaccination: number analyzed (Participants) | 8 | 8
  Serogroup Y: Before 12-13 months vaccination | 69.8 [11.0 to 441] | 20.7 [3.81 to 113]
  Serogroup W: 30 days after 3-month vaccination: number analyzed (Participants) | 4 | 6
  Serogroup W: 30 days after 3-month vaccination | 256 [NA to NA] — 95% CI was not computable as the sample size was too small to compute valid data. | 90.5 [5.16 to 1587]
  Serogroup W: Before 12-13 months vaccination: number analyzed (Participants) | 6 | 9
  Serogroup W: Before 12-13 months vaccination | 16.0 [1.40 to 183] | 4.67 [1.80 to 12.1]

42. Secondary Outcome: Percentage of Participants With rSBA Antibody Titers >=1:8 and >=1:128 Against Meningococcal Serogroups A, C, Y, and W - PPAS2
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by rSBA assay. Percentage of participants with rSBA antibody titers >=1:8 and >=1:128 for meningococcal serogroups A, C, Y, and W were reported in this outcome measure.
Time Frame: as for outcome 39
Population: as for outcome 41
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months)
Number analyzed (Participants) | 11 | 10
percentage of participants
  Serogroup A: 30 days after 3-month vaccination: >= 1:8: number analyzed (Participants) | 3 | 6
  Serogroup A: 30 days after 3-month vaccination: >= 1:8 | 66.7 [9.4 to 99.2] | 66.7 [22.3 to 95.7]
  Serogroup A: 30 days after 3-month vaccination: >= 1:128: number analyzed (Participants) | 3 | 6
  Serogroup A: 30 days after 3-month vaccination: >= 1:128 | 66.7 [9.4 to 99.2] | 16.7 [0.4 to 64.1]
  Serogroup A: Before 12-13 months vaccination: >= 1:8: number analyzed (Participants) | 7 | 9
  Serogroup A: Before 12-13 months vaccination: >= 1:8 | 42.9 [9.9 to 81.6] | 55.6 [21.2 to 86.3]
  Serogroup A: Before 12-13 months vaccination: >= 1:128: number analyzed (Participants) | 7 | 9
  Serogroup A: Before 12-13 months vaccination: >= 1:128 | 42.9 [9.9 to 81.6] | 44.4 [13.7 to 78.8]
  Serogroup C: 30 days after 3-month vaccination: >= 1:8: number analyzed (Participants) | 4 | 6
  Serogroup C: 30 days after 3-month vaccination: >= 1:8 | 100 [39.8 to 100] | 100 [54.1 to 100]
  Serogroup C: 30 days after 3-month vaccination: >= 1:128: number analyzed (Participants) | 4 | 6
  Serogroup C: 30 days after 3-month vaccination: >= 1:128 | 100 [39.8 to 100] | 83.3 [35.9 to 99.6]
  Serogroup C: Before 12-13 months vaccination: >= 1:8: number analyzed (Participants) | 8 | 9
  Serogroup C: Before 12-13 months vaccination: >= 1:8 | 87.5 [47.3 to 99.7] | 55.6 [21.2 to 86.3]
  Serogroup C: Before 12-13 months vaccination: >= 1:128: number analyzed (Participants) | 8 | 9
  Serogroup C: Before 12-13 months vaccination: >= 1:128 | 37.5 [8.5 to 75.5] | 11.1 [0.3 to 48.2]
  Serogroup Y: 30 days after 3-month vaccination: >= 1:8: number analyzed (Participants) | 3 | 6
  Serogroup Y: 30 days after 3-month vaccination: >= 1:8 | 100 [29.2 to 100] | 100 [54.1 to 100]
  Serogroup Y: 30 days after 3-month vaccination: >= 1:128: number analyzed (Participants) | 3 | 6
  Serogroup Y: 30 days after 3-month vaccination: >= 1:128 | 100 [29.2 to 100] | 50.0 [11.8 to 88.2]
  Serogroup Y: Before 12-13 months vaccination: >= 1:8: number analyzed (Participants) | 8 | 8
  Serogroup Y: Before 12-13 months vaccination: >= 1:8 | 87.5 [47.3 to 99.7] | 62.5 [24.5 to 91.5]
  Serogroup Y: Before 12-13 months vaccination: >= 1:128: number analyzed (Participants) | 8 | 8
  Serogroup Y: Before 12-13 months vaccination: >= 1:128 | 37.5 [8.5 to 75.5] | 25.0 [3.2 to 65.1]
  Serogroup W: 30 days after 3-month vaccination: >= 1:8: number analyzed (Participants) | 4 | 6
  Serogroup W: 30 days after 3-month vaccination: >= 1:8 | 100 [39.8 to 100] | 66.7 [22.3 to 95.7]
  Serogroup W: 30 days after 3-month vaccination: >= 1:128: number analyzed (Participants) | 4 | 6
  Serogroup W: 30 days after 3-month vaccination: >= 1:128 | 100 [39.8 to 100] | 66.7 [22.3 to 95.7]
  Serogroup W: Before 12-13 months vaccination: >= 1:8: number analyzed (Participants) | 6 | 9
  Serogroup W: Before 12-13 months vaccination: >= 1:8 | 50.0 [11.8 to 88.2] | 33.3 [7.5 to 70.1]
  Serogroup W: Before 12-13 months vaccination: >= 1:128: number analyzed (Participants) | 6 | 9
  Serogroup W: Before 12-13 months vaccination: >= 1:128 | 33.3 [4.3 to 77.7] | 0 [0 to 33.6]

43. Secondary Outcome: Number of Participants With Solicited Injection Site Reactions After Any Vaccination
Description: A solicited reaction (SR) was defined as an "expected" adverse reaction (AR) (sign or symptom) observed and reported under the conditions (nature and onset) pre-listed (i.e., solicited) in the protocol and case report form (CRF) and considered as related to vaccination. Solicited injection site reactions included injection site tenderness, injection site erythema, and injection site swelling and were planned to be collected and reported for each vaccine separately; and not planned to be collected for Rotavirus vaccine as the vaccine was administered orally, and no injection site reactions were expected to occur. Reported AEs for each arm were presented as pre-specified in the study protocol. Here, '0' in number analyzed field for MenACYW categories signifies that no participant was evaluable because in Group 3 MenACYW vaccine was not administered.
Time Frame: Within 7 days post any vaccination
Population: Analysis was performed on safety analysis set. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months) | Group 3: Bexsero® (2, 4, and 12 to 13 Months)
Number analyzed (Participants) | 314 | 314 | 157
Participants
  MenACYW conjugate vaccine: Tenderness: number analyzed (Participants) | 309 | 309 | 0
  MenACYW conjugate vaccine: Tenderness | 198 | 161 |
  MenACYW conjugate vaccine: Erythema: number analyzed (Participants) | 309 | 309 | 0
  MenACYW conjugate vaccine: Erythema | 220 | 205 |
  MenACYW conjugate vaccine: Swelling: number analyzed (Participants) | 309 | 309 | 0
  MenACYW conjugate vaccine: Swelling | 139 | 111 |
  Bexsero: Tenderness: number analyzed (Participants) | 310 | 312 | 155
  Bexsero: Tenderness | 266 | 230 | 138
  Bexsero: Erythema: number analyzed (Participants) | 310 | 312 | 155
  Bexsero: Erythema | 271 | 246 | 136
  Bexsero: Swelling: number analyzed (Participants) | 310 | 312 | 155
  Bexsero: Swelling | 234 | 192 | 118
  Infanrix hexa: Tenderness: number analyzed (Participants) | 309 | 312 | 155
  Infanrix hexa: Tenderness | 220 | 216 | 119
  Infanrix hexa: Erythema: number analyzed (Participants) | 309 | 312 | 155
  Infanrix hexa: Erythema | 254 | 231 | 117
  Infanrix hexa: Swelling: number analyzed (Participants) | 309 | 312 | 155
  Infanrix hexa: Swelling | 188 | 189 | 86
  Prevnar 13: Tenderness: number analyzed (Participants) | 309 | 312 | 155
  Prevnar 13: Tenderness | 195 | 196 | 118
  Prevnar 13: Erythema: number analyzed (Participants) | 309 | 311 | 155
  Prevnar 13: Erythema | 214 | 202 | 104
  Prevnar 13: Swelling: number analyzed (Participants) | 309 | 311 | 155
  Prevnar 13: Swelling | 140 | 137 | 69

44. Secondary Outcome: Number of Participants With Solicited Systemic Reactions After Any Vaccination
Description: A SR was an expected AR (sign or symptom) observed and reported under the conditions (nature and onset) prelisted (i.e., solicited) in the CRB and considered as related to the product administered. Solicited systemic reactions included fever, vomiting, crying abnormal, drowsiness, appetite lost, and irritability. Reported AEs for each arm were presented as pre-specified in the study protocol.
Time Frame: Within 7 days after any vaccination
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months) | Group 3: Bexsero® (2, 4, and 12 to 13 Months)
Number analyzed (Participants) | 314 | 314 | 157
Participants
  Fever: number analyzed (Participants) | 309 | 312 | 155
  Fever | 100 | 86 | 50
  Vomiting: number analyzed (Participants) | 310 | 312 | 155
  Vomiting | 173 | 172 | 71
  Crying abnormal: number analyzed (Participants) | 310 | 312 | 155
  Crying abnormal | 293 | 273 | 141
  Drowsiness: number analyzed (Participants) | 310 | 312 | 155
  Drowsiness | 275 | 275 | 137
  Appetite lost: number analyzed (Participants) | 310 | 312 | 155
  Appetite lost | 230 | 230 | 121
  Irritability: number analyzed (Participants) | 310 | 312 | 155
  Irritability | 306 | 299 | 147

ADVERSE EVENTS:
Time Frame: Unsolicited AEs: before first vaccination at the age of 3 months up to 30 days post any vaccination. SRs: within 7 days post any vaccination. Serious AEs: before first vaccination at the age of 3 months up to 30 days post last vaccination in each group (i.e., up to the age of 13 to 14 months)
Description: SR was an "expected" AR (sign or symptom) observed & reported under conditions (nature & onset) pre-listed in the protocol and CRF. Unsolicited AE: observed AE that does not fulfill the conditions prelisted in the CRF. Safety analysis set. Reported AEs for each arm were presented as pre-specified in protocol. In AE section, solicited reactions Fever, Crying abnormal, Drowsiness, and Appetite lost are reported under Pyrexia, Crying, Somnolence, and decreased appetite, respectively.
Arm/Group | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months) | Group 3: Bexsero® (2, 4, and 12 to 13 Months)
All-Cause Mortality (participants affected / at risk) | 0/314 | 0/314 | 0/157
Serious Adverse Events (participants affected / at risk) | 18/314 | 34/314 | 7/157
Other Adverse Events (participants affected / at risk) | 310/314 | 310/314 | 155/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) (N=314) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months) (N=314) | Group 3: Bexsero® (2, 4, and 12 to 13 Months) (N=157)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cystic Lymphangioma (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 0 (0)
Anaphylactic Reaction (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
Bronchiolitis (Infections and infestations) | 3 (3) | 4 (5) | 3 (3)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Herpes Virus Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Lymph Node Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia Viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Respiratory Syncytial Virus Bronchiolitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Respiratory Tract Infection Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral Rash (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Failure To Thrive (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Weight Gain Poor (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Embolic Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile Convulsion (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Head Titubation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cyanosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine + Bexsero® (2, 4, and 12 to 13 Months) (N=314) | Group 2: MenACYW Conjugate Vaccine + Bexsero® (2 and 4 Months) (N=314) | Group 3: Bexsero® (2, 4, and 12 to 13 Months) (N=157)
Constipation (Gastrointestinal disorders) | 12 (13) | 16 (16) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 42 (46) | 32 (42) | 23 (26)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 18 (19) | 14 (16) | 7 (8)
Teething (Gastrointestinal disorders) | 112 (195) | 115 (184) | 62 (98)
Vomiting (Gastrointestinal disorders) | 177 (323) | 174 (291) | 72 (144) — Vomiting events that occurred after 7 days post-vaccination were considered as unsolicited AEs.
Crying (General disorders) | 294 (820) | 274 (709) | 141 (418) — Crying/Crying abnormal events that occurred after 7 days post-vaccination were considered as unsolicited AEs.
Injection Site Bruising (General disorders) | 92 (154) | 89 (137) | 35 (64)
Injection Site Erythema (General disorders) | 294 (1806) | 281 (1455) | 144 (685)
Injection Site Mass (General disorders) | 26 (46) | 22 (40) | 14 (24)
Injection Site Pain (General disorders) | 277 (1521) | 263 (1295) | 141 (745)
Injection Site Swelling (General disorders) | 262 (1161) | 248 (909) | 127 (466)
Pyrexia (General disorders) | 115 (157) | 105 (137) | 58 (77) — Pyrexia/Fever events that occurred after 7 days post-vaccination were considered as unsolicited AEs.
Conjunctivitis (Infections and infestations) | 16 (16) | 11 (11) | 2 (2)
Nasopharyngitis (Infections and infestations) | 66 (98) | 56 (75) | 29 (39)
Upper Respiratory Tract Infection (Infections and infestations) | 35 (40) | 37 (51) | 11 (15)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 18 (20) | 19 (22) | 4 (5)
Decreased Appetite (Metabolism and nutrition disorders) | 230 (443) | 230 (425) | 121 (239)
Somnolence (Nervous system disorders) | 275 (688) | 275 (636) | 137 (320)
Irritability (Psychiatric disorders) | 306 (999) | 299 (905) | 147 (472)
Cough (Respiratory, thoracic and mediastinal disorders) | 30 (35) | 37 (43) | 9 (11)
Eczema (Skin and subcutaneous tissue disorders) | 10 (10) | 12 (14) | 9 (9)
Rash (Skin and subcutaneous tissue disorders) | 20 (23) | 30 (33) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT03632720/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/20/NCT03632720/SAP_001.pdf